CLINICAL TRIAL: NCT01235949
Title: Impact of Immediate or Delayed Prophylactic Antipyretic Treatment on the Immunogenicity, Reactogenicity and Safety of GlaxoSmithKline Biologicals' Pneumococcal Vaccine 1024850A and the Co-administered DTPa-combined Vaccines
Brief Title: Primary and Booster Vaccination Study With Pneumococcal Vaccine GSK1024850A and Prophylactic Antipyretic Treatment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 112921; 2010-019761-28 (EudraCT Number)
Record Dates: First submitted 2010-11-04; First posted 2010-11-08 (Estimated); Results first posted 2019-01-31 (Actual); Last update posted 2019-05-10 (Actual); Status verified 2019-04

CONDITIONS: Infections, Streptococcal
Keywords: Pneumococcal vaccine; Immunogenicity; Safety; Fever; Primary vaccination; Booster vaccination; Pneumococcal disease; Prophylactic antipyretic
MeSH Terms: conditions — Streptococcal Infections; Fever; Pneumococcal Infections | interventions — diphtheria-tetanus-acellular pertussis-inactivated poliovirus-Haemophilus influenzae b conjugate-hepatitis B vaccine; Ibuprofen; Acetaminophen

ARMS (18):
- Group IIBU (Experimental): Immediate ibuprofen group: subjects receiving immediate ibuprofen treatment after each primary vaccine dose
  Interventions: Biological: GSK1024850A (SynflorixTM); Biological: Infanrix hexa; Biological: Infanrix-IPV/Hib; Drug: Ibuprofen
- Group DIBU (Active Comparator): Delayed ibuprofen group: subjects receiving delayed ibuprofen treatment after each primary vaccine dose
  Interventions: Biological: GSK1024850A (SynflorixTM); Biological: Infanrix hexa; Biological: Infanrix-IPV/Hib; Drug: Ibuprofen
- Group NIBU (Active Comparator): No ibuprofen group: subjects receiving no prophylactic ibuprofen treatment after each primary vaccine dose
  Interventions: Biological: GSK1024850A (SynflorixTM); Biological: Infanrix hexa; Biological: Infanrix-IPV/Hib
- Group IPARA (Experimental): Immediate paracetamol group: subjects receiving immediate paracetamol treatment after each primary vaccine dose
  Interventions: Biological: GSK1024850A (SynflorixTM); Biological: Infanrix hexa; Biological: Infanrix-IPV/Hib; Drug: Paracetamol
- Group DPARA (Experimental): Delayed paracetamol group: subjects receiving delayed paracetamol treatment after each primary vaccine dose
  Interventions: Biological: GSK1024850A (SynflorixTM); Biological: Infanrix hexa; Biological: Infanrix-IPV/Hib; Drug: Paracetamol
- Group NPARA (Active Comparator): No paracetamol group: subjects receiving no prophylactic paracetamol treatment after each primary vaccine dose
  Interventions: Biological: GSK1024850A (SynflorixTM); Biological: Infanrix hexa; Biological: Infanrix-IPV/Hib
- Group IIBU-IIBU (Experimental): 1/3 of the subjects from the primary IIBU group receiving immediate ibuprofen treatment after booster vaccination
  Interventions: Biological: GSK1024850A (SynflorixTM); Biological: Infanrix hexa; Biological: Infanrix-IPV/Hib; Drug: Ibuprofen
- Group IIBU-DIBU (Experimental): 1/3 of the subjects from the primary IIBU group receiving delayed ibuprofen treatment after booster vaccination
  Interventions: Biological: GSK1024850A (SynflorixTM); Biological: Infanrix hexa; Biological: Infanrix-IPV/Hib
- Group IIBU-NIBU (Experimental): 1/3 of the subjects from the primary IIBU group receiving no prophylactic ibuprofen treatment after booster vaccination
  Interventions: Biological: GSK1024850A (SynflorixTM); Biological: Infanrix hexa; Biological: Infanrix-IPV/Hib; Drug: Ibuprofen
- Group DIBU-IIBU (Experimental): 1/3 of the subjects from the primary DIBU group receiving immediate ibuprofen treatment after booster vaccination
  Interventions: Biological: GSK1024850A (SynflorixTM); Biological: Infanrix hexa; Biological: Infanrix-IPV/Hib; Drug: Ibuprofen
- Group DIBU-DIBU (Experimental): 1/3 of the subjects from the primary DIBU group receiving delayed ibuprofen treatment after booster vaccination
  Interventions: Biological: GSK1024850A (SynflorixTM); Biological: Infanrix hexa; Biological: Infanrix-IPV/Hib; Drug: Ibuprofen
- Group DIBU-NIBU (Experimental): 1/3 of the subjects from the primary DIBU group receiving no prophylactic ibuprofen treatment after booster vaccination
  Interventions: Biological: GSK1024850A (SynflorixTM); Biological: Infanrix hexa; Biological: Infanrix-IPV/Hib
- Group NIBU-IIBU (Experimental): 1/3 of the subjects from the primary NIBU group receiving immediate ibuprofen treatment after booster vaccination
  Interventions: Biological: GSK1024850A (SynflorixTM); Biological: Infanrix hexa; Biological: Infanrix-IPV/Hib; Drug: Ibuprofen
- Group NIBU-DIBU (Experimental): 1/3 of the subjects from the primary NIBU group receiving delayed ibuprofen treatment after booster vaccination
  Interventions: Biological: GSK1024850A (SynflorixTM); Biological: Infanrix hexa; Biological: Infanrix-IPV/Hib; Drug: Ibuprofen
- Group NIBU-NIBU (Active Comparator): 1/3 of the subjects from the primary NIBU group receiving no prophylactic ibuprofen treatment after booster vaccination
  Interventions: Biological: GSK1024850A (SynflorixTM); Biological: Infanrix hexa; Biological: Infanrix-IPV/Hib
- Group IPARA-NPARA (Experimental): subjects from the primary IPARA group receiving no paracetamol treatment after booster vaccination
  Interventions: Biological: GSK1024850A (SynflorixTM); Biological: Infanrix hexa; Biological: Infanrix-IPV/Hib
- Group DPARA-IPARA (Experimental): subjects from the primary DPARA group receiving immediate paracetamol treatment after booster vaccination
  Interventions: Biological: GSK1024850A (SynflorixTM); Biological: Infanrix hexa; Biological: Infanrix-IPV/Hib; Drug: Paracetamol
- Group NPARA-IPARA (Experimental): subjects from the primary NPARA group receiving immediate paracetamol treatment after booster vaccination
  Interventions: Biological: GSK1024850A (SynflorixTM); Biological: Infanrix hexa; Biological: Infanrix-IPV/Hib; Drug: Paracetamol

INTERVENTIONS:
Biological: GSK1024850A (SynflorixTM) — Intramuscular injection, 4 doses
Biological: Infanrix hexa — Intramuscular injection, 3 doses
Biological: Infanrix-IPV/Hib — Intramuscular injection, 1 dose
Drug: Ibuprofen — Oral administration, 3 doses in the 24 hours following vaccination with an interval of 6-8 hours between doses and with dosage based on the subject's body weight
  Other Names: Nurofen for Children
  Arms: Group DIBU; Group DIBU-DIBU; Group DIBU-IIBU; Group IIBU; Group IIBU-IIBU; Group IIBU-NIBU; Group NIBU-DIBU; Group NIBU-IIBU
Drug: Paracetamol — Oral administration, 3 doses in the 24 hours following vaccination with an interval of 6-8 hours between doses and with dosage based on the subject's body weight
  Other Names: Panadol Baby
  Arms: Group DPARA; Group DPARA-IPARA; Group IPARA; Group NPARA-IPARA

SUMMARY:
The aim of the current study is to determine whether ibuprofen, given as immediate or delayed prophylactic antipyretic treatment in a standardized manner, significantly impacts the immune response in children receiving primary vaccination with GlaxoSmithKline (GSK) Biologicals' 10-valent pneumococcal conjugate vaccine, co-administered with DTPa-combined vaccines, at 3, 4 and 5 months of age.

In addition, this study will further evaluate the impact of prophylactic administration of paracetamol following primary vaccination with immediate or delayed administration or when given in an immediate manner at the time of the booster dose.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that their parent(s)/Legally Acceptable Representative(s) (LAR) can and will comply with the requirements of the protocol.
* A male or female between, and including, 12 and 16 weeks (84-118 days) of age at the time of the first vaccination.
* Written informed consent obtained from the parent(s)/LAR(s) of the subject.
* Free of obvious health problems as established by medical history and clinical examination before entering into the study.
* Born after a gestation period of 36 to 42 weeks inclusive.

Exclusion Criteria:

* Use of any investigational or non-registered product other than the study vaccines/products within 30 days preceding the first dose of study vaccine/product, or planned use during the study period.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product (.
* Indication, other than specified in the protocol, for prophylactic or therapeutic antipyretic treatment during the study period.
* Treatment with antipyretics in the 24 hours before study vaccination or planned administration of antipyretics in the 24 hours after study vaccination.
* Chronic administration of immunosuppressants or other immune-modifying drugs since birth.
* Planned administration/administration of a vaccine not foreseen by the study protocol during the period starting 30 days before each dose of study vaccine and ending 30 days after with the exception of locally recommended (pandemic) influenza vaccines, and those should be documented in the eCRF.
* Previous vaccination against diphtheria, tetanus, pertussis, polio, hepatitis B, Haemophilus influenzae type b and/or Streptococcus pneumoniae with the exception of the vaccines where the first dose may be given within the first two weeks of life according to the national recommendations.
* History of intercurrent diphtheria, tetanus, pertussis, polio, hepatitis B, Haemophilus influenzae type b disease.
* History of any allergic disease or reaction likely to be exacerbated by any component of the vaccines or prophylactic antipyretic treatment, i.e. ibuprofen or paracetamol, as specified in the protocol.
* History of any seizures or progressive neurological disease.
* Acute disease and/or fever at the time of enrolment. The study entry should be delayed until the illness has improved.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination .
* A family history of congenital or hereditary immunodeficiency.
* Major congenital defects or serious chronic illness.
* Administration of immunoglobulins and/or any blood products since birth or planned administration during entire study period.
* Any contraindication to treatment with ibuprofen as described in the ibuprofen summary of product characteristics (SPC).
* Any contraindication to treatment with paracetamol as described in the paracetamol SPC.
* Body weight < 5 kg at the time of enrolment.
* Child in care.

Ages: 12 Weeks to 16 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 850 (Actual)
Dates: Start 2010-11-12 (Actual); Primary Completion 2012-03-28 (Actual); Study Completion 2012-12-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (12):
- Romania (12):
  - GSK Investigational Site, Bacau
  - GSK Investigational Site, Brasov
  - GSK Investigational Site, Brăila
  - GSK Investigational Site, Bucharest
  - GSK Investigational Site, Călăraşi
  - GSK Investigational Site, Cluj-Napoca
  - GSK Investigational Site, Constanța
  - GSK Investigational Site, Galati
  - GSK Investigational Site, Iași
  - GSK Investigational Site, Pantelimon
  - GSK Investigational Site, Sibiu
  - GSK Investigational Site, Timișoara

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Falup-Pecurariu O, Man SC, Neamtu ML, Chicin G, Baciu G, Pitic C, Cara AC, Neculau AE, Burlea M, Brinza IL, Schnell CN, Sas V, Lupu VV, Francois N, Swinnen K, Borys D. Effects of prophylactic ibuprofen and paracetamol administration on the immunogenicity and reactogenicity of the 10-valent pneumococcal non-typeable Haemophilus influenzae protein D conjugated vaccine (PHiD-CV) co-administered with DTPa-combined vaccines in children: An open-label, randomized, controlled, non-inferiority trial. Hum Vaccin Immunother. 2017 Mar 4;13(3):649-660. doi: 10.1080/21645515.2016.1223001. Epub 2016 Aug 19. PMID 27541270
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: 112921 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 112921 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 112921 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 112921 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 112921 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 112921 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Among the 850 subjects enrolled in the study, 35 subjects were excluded for lack of confidence in the integrity of the data and 3 subjects were allocated with subject number but didn't receive any vaccination.
Pre-assignment Details: During the screening the following steps occurred: check for inclusion/exclusion criteria, contraindications/precautions, medical history of the subjects and signing informed consent forms.
Groups:
- IIBU Group: Healthy male and female subjects between and including 12 and 16 weeks of age, who received immediate ibuprofen (IIBU) administration with Nurofen™ for Children after each primary vaccination dose of Synflorix™ vaccine at 3, 4 and 5 months of age, co-administered with Infanrix hexa™ at 3 and 5 months of age and with Infanrix™-IPV/Hib at 4 months of age. For immediate oral administration of Nurofen™: antipyretic dose 1 was administered at the time of vaccination, antipyretic doses 2 and 3 were administered 6-8 hours after the previous dose of antipyretic. All three vaccines were administered intramuscularly into the right or left thigh. This group is applicable for all analysis related to the primary phase of the study as well as for Serious Adverse Event (SAE) follow-up for the entire study period.
- DIBU Group: Healthy male and female subjects between and including 12 and 16 weeks of age, who received delayed ibuprofen (DIBU) administration with Nurofen™ for Children after each primary vaccination dose of Synflorix™ vaccine at 3, 4 and 5 months of age, co-administered with Infanrix hexa™ at 3 and 5 months of age and with Infanrix™-IPV/Hib at 4 months of age. For delayed oral administration of Nurofen™: antipyretic dose 1 was administered 4-6 hours after vaccination, antipyretic doses 2 and 3 were administered 6-8 hours after the previous dose of antipyretic. All three vaccines were administered intramuscularly into the right or left thigh. This group is applicable for all analysis related to the primary phase of the study as well as for SAE follow-up for the entire study period.
- NIBU Group: Healthy male and female subjects between and including 12 and 16 weeks of age, who received no prophylactic ibuprofen (NIBU) administration after each primary vaccination dose of Synflorix™ vaccine at 3, 4 and 5 months of age, co-administered with Infanrix hexa™ at 3 and 5 months of age and with Infanrix™-IPV/Hib at 4 months of age. All three vaccines were administered intramuscularly into the right or left thigh. This group is applicable for all analysis related to the primary phase of the study as well as for SAE follow-up for the entire study period.
- IPARA Group: Healthy male and female subjects between and including 12 and 16 weeks of age, who received immediate paracetamol (IPARA) administration with Panadol™ Baby after each primary vaccination dose of Synflorix™ vaccine at 3, 4 and 5 months of age, co-administered with Infanrix hexa™ at 3 and 5 months of age and with Infanrix™-IPV/Hib at 4 months of age. For immediate oral administration of Panadol™: antipyretic dose 1 was administered at the time of vaccination, antipyretic doses 2 and 3 were administered 6-8 hours after the previous dose of antipyretic. All three vaccines were administered intramuscularly into the right or left thigh. This group is applicable for all analysis related to the primary phase of the study as well as for SAE follow-up for the entire study period.
- DPARA Group: Healthy male and female subjects between and including 12 and 16 weeks of age, who received delayed paracetamol (DPARA) administration with Panadol™ Baby after each primary vaccination dose of Synflorix™ vaccine at 3, 4 and 5 months of age, co-administered with Infanrix hexa™ at 3 and 5 months of age and with Infanrix™-IPV/Hib at 4 months of age. For delayed oral administration of Panadol™: antipyretic dose 1 was administered 4-6 hours after vaccination, antipyretic doses 2 and 3 were administered 6-8 hours after the previous dose of antipyretic. All three vaccines were administered intramuscularly into the right or left thigh. This group is applicable for all analysis related to the primary phase of the study as well as for SAE follow-up for the entire study period.
- NPARA Group: Healthy male and female subjects between and including 12 and 16 weeks of age, who received no prophylactic paracetamol (NPARA) administration after each primary vaccination dose of Synflorix™ vaccine at 3, 4 and 5 months of age, co-administered with Infanrix hexa™ at 3 and 5 months of age and with Infanrix™-IPV/Hib at 4 months of age. All three vaccines were administered intramuscularly into the right or left thigh. This group is applicable for all analysis related to the primary phase of the study as well as for SAE follow-up for the entire study period.
- IIBU-IIBU Group: 1/3 of the subjects from the primary Synflorix/Immediate Ibuprofen Group (IIBU Group) received immediate ibuprofen treatment (IIBU) with Nurofen™ for Children after booster vaccination with Synflorix™ vaccine co-administered with Infanrix hexa™ vaccine at 12-15 months of age. For immediate oral administration of Nurofen™: antipyretic dose 1 was administered at the time of vaccination, antipryretic doses 2 and 3 were administered 6-8 hours after the previous dose of antipyretic. Both vaccines were administered intramuscularly into the right/left thigh or into the deltoid muscle.
- IIBU-DIBU Group: 1/3 of the subjects from the primary Synflorix/Immediate Ibuprofen Group (IIBU Group) received delayed ibuprofen treatment (DIBU) with Nurofen™ for Children after booster vaccination with Synflorix™ vaccine co-administered with Infanrix hexa™ vaccine at 12-15 months of age. For delayed oral administration of Nurofen™: antipyretic dose 1 was administered 4-6 hours after vaccination, antipyretic doses 2 and 3 were administered 6-8 hours after the previous dose of antipyretic. Both vaccines were administered intramuscularly into the right/left thigh or into the deltoid muscle.
- IIBU-NIBU Group: 1/3 of the subjects from the primary Synflorix/Immediate Ibuprofen Group (IIBU Group) received no prophylactic ibuprofen treatment (NIBU) with Nurofen™ for Children after the booster vaccination with Synflorix™ vaccine co-administered with Infanrix hexa™ vaccine at 12-15 months of age. Both vaccines were administered intramuscularly into the right/left thigh or into the deltoid muscle.
- DIBU-IIBU Group: 1/3 of the subjects from the primary Synflorix/Delayed Ibuprofen Group (DIBU Group) received immediate ibuprofen treatment (IIBU) with Nurofen™ for Children after booster vaccination with Synflorix™ vaccine co-administered with Infanrix hexa™ vaccine at 12-15 months of age. For immediate oral administration of Nurofen™: antipyretic dose 1 was administered at the time of vaccination, antipyretic doses 2 and 3 were administered 6-8 hours after the previous dose of antipyretic. Both vaccines were administered intramuscularly into the right/left thigh or into the deltoid muscle.
- DIBU-DIBU Group: 1/3 of the subjects from the primary Synflorix/Delayed Ibuprofen Group (DIBU Group) received delayed ibuprofen treatment (DIBU) with Nurofen™ for Children after booster vaccination with Synflorix™ vaccine co-administered with Infanrix hexa™ vaccine at 12-15 months of age. For delayed oral administration of Nurofen™: antipyretic dose 1 was administered 4-6 hours after vaccination, antipyretic doses 2 and 3 were administered 6-8 hours after the previous dose of antipyretic. Both vaccines were administered intramuscularly into the right/left thigh or into the deltoid muscle.
- DIBU-NIBU Group: 1/3 of the subjects from the primary Synflorix/Delayed Ibuprofen Group (DIBU Group) received no prophylactic ibuprofen treatment (NIBU) with Nurofen™ for Children after the booster vaccination with Synflorix™ vaccine co-administered with Infanrix hexa™ vaccine at 12-15 months of age. Both vaccines were administered intramuscularly into the right/left thigh or into the deltoid muscle.
- NIBU-IIBU Group: 1/3 of the subjects from the primary Synflorix/No Ibuprofen Group (NIBU Group) received immediate ibuprofen treatment (IIBU) with Nurofen™ for Children after booster vaccination with Synflorix™ vaccine co-administered with Infanrix hexa™ vaccine at 12-15 months of age. For immediate oral administration of Nurofen™: antipyretic dose 1 was administered at the time of vaccination, antipyretic doses 2 and 3 were administered 6-8 hours after the previous dose of antipyretic. Both vaccines were administered intramuscularly into the right/left thigh or into the deltoid muscle.
- NIBU-DIBU Group: 1/3 of the subjects from the primary Synflorix/No Ibuprofen Group (DIBU Group) received delayed ibuprofen treatment (DIBU) with Nurofen™ for Children after booster vaccination with Synflorix™ vaccine co-administered with Infanrix hexa™ vaccine at 12-15 months of age. For delayed oral administration of Nurofen™: antipyretic dose 1 was administered 4-6 hours after vaccination, antipyretic doses 2 and 3 were administered 6-8 hours after the previous dose of antipyretic. Both vaccines were administered intramuscularly into the right/left thigh or into the deltoid muscle.
- NIBU-NIBU Group: 1/3 of the subjects from the primary Synflorix/No Ibuprofen Group (DIBU Group) received no prophylactic ibuprofen treatment (NIBU) with Nurofen™ for Children after the booster vaccination with Synflorix™ vaccine co-administered with Infanrix hexa™ vaccine at 12-15 months of age. Both vaccines were administered intramuscularly into the right/left thigh or into the deltoid muscle.
- IPARA-NPARA Group: Subjects from the primary Synflorix/Immediate Paracetamol Group (IPARA Group) received no prophylactic paracetamol treatment (NPARA) with Panadol™ Baby after the booster vaccination with Synflorix™ vaccine co-administered with Infanrix hexa™ vaccine at 12-15 months of age. Both vaccines were administered intramuscularly into the right/left thigh or into the deltoid muscle.
- DPARA-IPARA Group: Subjects from the primary Synflorix/Delayed Paracetamol Group (DPARA Group) received immediate paracetamol treatment (IPARA) with Panadol™ Baby after booster vaccination with Synflorix™ vaccine co-administered with Infanrix hexa™ vaccine at 12-15 months of age. For immediate oral administration of Panadol™: antipyretic dose 1 was administered at the time of vaccination, antipyretic doses 2 and 3 were administered 6-8 hours after the previous dose of antipyretic. Both vaccines were administered intramuscularly into the right/left thigh or into the deltoid muscle.
- NPARA-IPARA Group: Subjects from the primary Synflorix/No Paracetamol Group (NPARA Group) received immediate paracetamol treatment (IPARA) with Panadol™ Baby after booster vaccination with Synflorix™ vaccine co-administered with Infanrix hexa™ vaccine at 12-15 months of age. For immediate oral administration of Panadol™: antipyretic dose 1 was administered at the time of vaccination, antipyretic doses 2 and 3 were administered 6-8 hours after the previous dose of antipyretic. Both vaccines were administered intramuscularly into the right/left thigh or into the deltoid muscle.
Period: Primary Phase
Arm/Group | IIBU Group | DIBU Group | NIBU Group | IPARA Group | DPARA Group | NPARA Group | IIBU-IIBU Group | IIBU-DIBU Group | IIBU-NIBU Group | DIBU-IIBU Group | DIBU-DIBU Group | DIBU-NIBU Group | NIBU-IIBU Group | NIBU-DIBU Group | NIBU-NIBU Group | IPARA-NPARA Group | DPARA-IPARA Group | NPARA-IPARA Group
Started | 198 | 198 | 199 | 71 | 72 | 74 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 194 (After Primary Phase completion, 7 subjects were not willing to participate in the Booster Phase) | 195 (After Primary Phase completion, 6 subjects were not willing to participate in the Booster Phase) | 196 (After Primary Phase completion, 6 subjects were not willing to participate in the Booster Phase) | 69 (After Primary Phase completion, 2 subjects were not willing to participate in the Booster Phase) | 71 (After Primary Phase completion, 3 subjects were not willing to participate in the Booster Phase) | 67 (After Primary Phase completion, all subjects were willing to participate in the Booster Phase) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 4 | 3 | 3 | 2 | 1 | 7 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Migrated/moved from study area | 1 | 1 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 2 | 2 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Booster Phase
Arm/Group | IIBU Group | DIBU Group | NIBU Group | IPARA Group | DPARA Group | NPARA Group | IIBU-IIBU Group | IIBU-DIBU Group | IIBU-NIBU Group | DIBU-IIBU Group | DIBU-DIBU Group | DIBU-NIBU Group | NIBU-IIBU Group | NIBU-DIBU Group | NIBU-NIBU Group | IPARA-NPARA Group | DPARA-IPARA Group | NPARA-IPARA Group
Started (After Primary Phase completion, 24 subjects were not willing to participate in the Booster Phase) | 0 (re-randomized to diverse treatments (IIBU-IIBU, IIBU-DIBU and IIBU-NIBU Groups) in booster phase) | 0 (re-randomized to diverse treatments (DIBU-IIBU, DIBU-DIBU and DIBU-NIBU Groups) in booster phase) | 0 (re-randomized to diverse treatments (NIBU-IIBU, NIBU-DIBU and NIBU-NIBU Groups) in booster phase) | 0 (subjects re-randomized to IPARA-NPARA Group in booster phase) | 0 (subjects re-randomized to DPARA-IPARA Group in booster phase) | 0 (subjects re-randomized to NPARA-IPARA Group in booster phase) | 64 (1/3 of subjects from primary IIBU group re-randomized to receive diverse booster phase treatments) | 60 (1/3 of subjects from primary IIBU group re-randomized to receive diverse booster phase treatments) | 63 (1/3 of subjects from primary IIBU group re-randomized to receive diverse booster phase treatments) | 63 (1/3 of subjects from primary DIBU group re-randomized to receive diverse booster phase treatments) | 63 (1/3 of subjects from primary DIBU group re-randomized to receive diverse booster phase treatments) | 63 (1/3 of subjects from primary DIBU group re-randomized to receive diverse booster phase treatments) | 63 (1/3 of subjects from primary NIBU group re-randomized to receive diverse booster phase treatments) | 65 (1/3 of subjects from primary NIBU group re-randomized to receive diverse booster phase treatments) | 62 (1/3 of subjects from primary NIBU group re-randomized to receive diverse booster phase treatments) | 67 (subjects from the primary IPARA group continuing in booster phase with different treatment) | 68 (subjects from the primary DPARA group continuing in booster phase with different treatment) | 67 (subjects from the primary NPARA group continuing in booster phase with different treatment)
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 64 | 59 | 61 | 62 | 61 | 60 | 60 | 65 | 60 | 66 | 68 | 65
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 2 | 3 | 3 | 0 | 2 | 1 | 0 | 2
Not completed — Migrated/moved from study area | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 2 | 0 | 2 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IIBU Group | DIBU Group | NIBU Group | IPARA Group | DPARA Group | NPARA Group | IIBU-IIBU Group | IIBU-DIBU Group | IIBU-NIBU Group | DIBU-IIBU Group | DIBU-DIBU Group | DIBU-NIBU Group | NIBU-IIBU Group | NIBU-DIBU Group | NIBU-NIBU Group | IPARA-NPARA Group | DPARA-IPARA Group | NPARA-IPARA Group | Total
Number analyzed (Participants) | 198 | 198 | 199 | 71 | 72 | 74 | 64 | 60 | 63 | 63 | 63 | 63 | 63 | 65 | 62 | 67 | 68 | 67 | 1580
Age, Continuous [Mean (Standard Deviation); unit: Weeks] — Primary Phase Groups Population: This baseline measure refers only to the primary phase groups.
  Weeks
    number analyzed (Participants) | 198 | 198 | 199 | 71 | 72 | 74 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 812
    (all) | 13.1 (1.15) | 13 (1.2) | 12.9 (1.14) | 13 (1.3) | 13.2 (1.3) | 13.2 (1.11) |  |  |  |  |  |  |  |  |  |  |  |  | 13.04 (1.18)
Age, Continuous [Mean (Standard Deviation); unit: Months] — Booster Phase Groups Population: This baseline measure refers only to the booster phase groups.
  Months
    number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 64 | 60 | 63 | 63 | 63 | 63 | 63 | 65 | 62 | 67 | 68 | 67 | 768
    (all) |  |  |  |  |  |  | 12.3 (0.64) | 12.2 (0.49) | 12.3 (0.57) | 12.2 (0.45) | 12.4 (0.63) | 12.4 (0.73) | 12.3 (0.63) | 12.3 (0.57) | 12.3 (0.70) | 12.3 (0.73) | 12.3 (0.56) | 12.4 (0.63) | 12.3 (0.61)
Sex: Female, Male [Count of Participants; unit: Participants] — Primary Phase Groups Population: This baseline measure refers only to the primary phase groups.
  Participants
    number analyzed (Participants) | 198 | 198 | 199 | 71 | 72 | 74 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 812
    Female | 90 | 86 | 104 | 39 | 40 | 38 |  |  |  |  |  |  |  |  |  |  |  |  | 397
    Male | 108 | 112 | 95 | 32 | 32 | 36 |  |  |  |  |  |  |  |  |  |  |  |  | 415
Sex: Female, Male [Count of Participants; unit: Participants] — Booster Phase Groups Population: This baseline measure refers only to the booster phase groups.
  Participants
    number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 64 | 60 | 63 | 63 | 63 | 63 | 63 | 65 | 62 | 67 | 68 | 67 | 768
    Female |  |  |  |  |  |  | 29 | 27 | 29 | 23 | 33 | 27 | 32 | 35 | 35 | 37 | 39 | 33 | 379
    Male |  |  |  |  |  |  | 35 | 33 | 34 | 40 | 30 | 36 | 31 | 30 | 27 | 30 | 29 | 34 | 389
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Primary Phase Groups Population: This baseline measure refers only to the primary phase groups.
  Participants
    White- Caucasian/European heritage: number analyzed (Participants) | 198 | 198 | 199 | 71 | 72 | 74 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 812
    White- Caucasian/European heritage | 198 | 197 | 198 | 70 | 72 | 72 |  |  |  |  |  |  |  |  |  |  |  |  | 807
    White - Arabic/North African Heritage: number analyzed (Participants) | 198 | 198 | 199 | 71 | 72 | 74 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 812
    White - Arabic/North African Heritage | 0 | 0 | 0 | 1 | 0 | 1 |  |  |  |  |  |  |  |  |  |  |  |  | 2
    Not specified: number analyzed (Participants) | 198 | 198 | 199 | 71 | 72 | 74 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 812
    Not specified | 0 | 1 | 1 | 0 | 0 | 1 |  |  |  |  |  |  |  |  |  |  |  |  | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Booster Phase Groups Population: This baseline measure refers only to the booster phase groups.
  Participants
    White- Caucasian/European heritage: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 64 | 60 | 63 | 63 | 63 | 63 | 63 | 65 | 62 | 67 | 68 | 67 | 768
    White- Caucasian/European heritage |  |  |  |  |  |  | 64 | 60 | 63 | 63 | 63 | 62 | 63 | 65 | 62 | 66 | 68 | 66 | 765
    White - Arabic/North African Heritage: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 64 | 60 | 63 | 63 | 63 | 63 | 63 | 65 | 62 | 67 | 68 | 67 | 768
    White - Arabic/North African Heritage |  |  |  |  |  |  | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
    Not specified: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 64 | 60 | 63 | 63 | 63 | 63 | 63 | 65 | 62 | 67 | 68 | 67 | 768
    Not specified |  |  |  |  |  |  | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Antibody Concentrations Against Vaccine Pneumococcal Serotypes Greater Than or Equal to (≥) the Cut-off
Description: Antibodies against the vaccine pneumococcal serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F (Anti-1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F) have been assessed by 22F-inhibition enzyme-linked immunosorbent assay (ELISA). The cut-off value of the assay was an antibody concentration greater than or equal to (≥) 0.2 micrograms per milliliter (μg/mL).
Time Frame: One month after primary immunization (At Month 3)
Population: The analysis was performed on the According-to-Protocol (ATP) cohort for immunogenicity, which included all evaluable subjects for whom immunogenicity data and assay results for antibodies against at least one study vaccine antigen component after vaccination were available.
Measure: Count of Participants; unit: Participants
Arm/Group | IIBU Group | DIBU Group | NIBU Group | IPARA Group | DPARA Group | NPARA Group
Number analyzed (Participants) | 154 | 158 | 164 | 55 | 55 | 56
Participants
  Anti-1: number analyzed (Participants) | 144 | 155 | 161 | 54 | 51 | 55
  Anti-1 | 144 | 155 | 160 | 52 | 50 | 55
  Anti-4: number analyzed (Participants) | 146 | 155 | 159 | 55 | 51 | 56
  Anti-4 | 145 | 155 | 158 | 53 | 51 | 56
  Anti-5: number analyzed (Participants) | 143 | 154 | 157 | 53 | 50 | 54
  Anti-5 | 143 | 154 | 156 | 53 | 50 | 54
  Anti-6B: number analyzed (Participants) | 144 | 155 | 157 | 53 | 51 | 55
  Anti-6B | 121 | 135 | 133 | 42 | 37 | 48
  Anti-7F: number analyzed (Participants) | 154 | 157 | 164 | 55 | 55 | 56
  Anti-7F | 153 | 157 | 164 | 55 | 55 | 56
  Anti-9V: number analyzed (Participants) | 145 | 153 | 157 | 53 | 50 | 54
  Anti-9V | 144 | 153 | 155 | 53 | 50 | 53
  Anti-14: number analyzed (Participants) | 144 | 154 | 155 | 53 | 50 | 53
  Anti-14 | 144 | 153 | 154 | 53 | 50 | 53
  Anti-18C: number analyzed (Participants) | 144 | 154 | 157 | 53 | 50 | 54
  Anti-18C | 143 | 153 | 155 | 52 | 50 | 54
  Anti-19F: number analyzed (Participants) | 145 | 154 | 158 | 53 | 50 | 54
  Anti-19F | 145 | 152 | 157 | 53 | 50 | 54
  Anti-23F: number analyzed (Participants) | 148 | 158 | 162 | 54 | 53 | 55
  Anti-23F | 136 | 141 | 149 | 47 | 43 | 50
Statistical Analysis 1: Comparison: IIBU Group vs NIBU Group; At one month after primary immunization, the difference between groups (NIBU minus IIBU), in terms of percentage of subjects with pneumococcal antibody concentrations ≥ 0.2 µg/mL were calculated for anti-pneumococccal serotype 1; Test type: Non-Inferiority — Criterion for evaluation of non-inferiority: The upper limit (UL) of the 2-sided 98.25% confidence interval (98.25% CI) (adjusted 1-sided alpha = 0.875%) of the difference between groups (NIBU minus IIBU), in terms of percentage of subjects with pneumococcal antibody concentrations ≥ 0.2 µg/mL, was lower than (<) 10% for at least 7 out of the 10 pneumococcal serotypes; Difference in percentages = -0.62, 98.25% CI 2-sided [-4.52 to 3.17]
Statistical Analysis 2: Comparison: IIBU Group vs NIBU Group; At one month after primary immunization, the difference between groups (NIBU minus IIBU), in terms of percentage of subjects with pneumococcal antibody concentrations ≥ 0.2 µg/mL were calculated for anti-pneumococcal serotype 4; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Difference in percentages = 0.06, 98.25% CI 2-sided [-3.94 to 4.38]
Statistical Analysis 3: Comparison: IIBU Group vs NIBU Group; At one month after primary immunization, the difference between groups (NIBU minus IIBU), in terms of percentage of subjects with pneumococcal antibody concentrations ≥ 0.2 µg/mL were calculated for anti-pneumococccal serotype 5; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Difference in percentages = -0.64, 98.25% CI 2-sided [-4.63 to 3.19]
Statistical Analysis 4: Comparison: IIBU Group vs NIBU Group; At one month after primary immunization, the difference between groups (NIBU minus IIBU), in terms of percentage of subjects with pneumococcal antibody concentrations ≥ 0.2 µg/mL were calculated for anti-pneumococccal serotype 6B; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Difference in percentages = 0.69, 98.25% CI 2-sided [-9.4 to 10.99]
Statistical Analysis 5: Comparison: IIBU Group vs NIBU Group; At one month after primary immunization, the difference between groups (NIBU minus IIBU), in terms of percentage of subjects with pneumococcal antibody concentrations ≥ 0.2 µg/mL were calculated for anti-pneumococccal serotype 7F; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Difference in percentages = 0.65, 98.25% CI 2-sided [-2.7 to 4.71]
Statistical Analysis 6: Comparison: IIBU Group vs NIBU Group; At one month after primary immunization, the difference between groups (NIBU minus IIBU), in terms of percentage of subjects with pneumococcal antibody concentrations ≥ 0.2 µg/mL were calculated for anti-pneumococccal serotype 9V; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Difference in percentages = -0.58, 98.25% CI 2-sided [-5.05 to 3.82]
Statistical Analysis 7: Comparison: IIBU Group vs NIBU Group; At one month after primary immunization, the difference between groups (NIBU minus IIBU), in terms of percentage of subjects with pneumococcal antibody concentrations ≥ 0.2 µg/mL were calculated for anti-pneumococccal serotype 14; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Difference in percentages = -0.65, 98.25% CI 2-sided [-4.68 to 3.15]
Statistical Analysis 8: Comparison: IIBU Group vs NIBU Group; At one month after primary immunization, the difference between groups (NIBU minus IIBU), in terms of percentage of subjects with pneumococcal antibody concentrations ≥ 0.2 µg/mL were calculated for anti-pneumococccal serotype 18C; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Difference in percentages = -0.58, 98.25% CI 2-sided [-5.04 to 3.85]
Statistical Analysis 9: Comparison: IIBU Group vs NIBU Group; At one month after primary immunization, the difference between groups (NIBU minus IIBU), in terms of percentage of subjects with pneumococcal antibody concentrations ≥ 0.2 µg/mL were calculated for anti-pneumococccal serotype 19F; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Difference in percentages = -0.63, 98.25% CI 2-sided [-4.6 to 3.14]
Statistical Analysis 10: Comparison: IIBU Group vs NIBU Group; At one month after primary immunization, the difference between groups (NIBU minus IIBU), in terms of percentage of subjects with pneumococcal antibody concentrations ≥ 0.2 µg/mL were calculated for anti-pneumococccal serotype 23F; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Difference in percentages = 0.08, 98.25% CI [-7.66 to 8.1]
Statistical Analysis 11: Comparison: DIBU Group vs NIBU Group; At one month after primary immunization, the difference between groups (NIBU minus DIBU), in terms of percentage of subjects with pneumococcal antibody concentrations ≥ 0.2 µg/mL were calculated for anti-pneumococccal serotype 1; Test type: Non-Inferiority — Criterion for evaluation of non-inferiority: The upper limit (UL) of the 2-sided 98.25% confidence interval (98.25% CI) (adjusted 1-sided alpha = 0.875%) of the difference between groups (NIBU minus DIBU), in terms of percentage of subjects with pneumococcal antibody concentrations ≥ 0.2 µg/mL, was lower than (<) 10% for at least 7 out of the 10 pneumococcal serotypes; Difference in percentages = -0.62, 98.25% CI 2-sided [-4.52 to 2.91]
Statistical Analysis 12: Comparison: DIBU Group vs NIBU Group; At one month after primary immunization, the difference between groups (NIBU minus DIBU), in terms of percentage of subjects with pneumococcal antibody concentrations ≥ 0.2 µg/mL were calculated for anti-pneumococccal serotype 4; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 11]; Difference in percentages = -0.63, 98.25% CI 2-sided [-4.57 to 2.91]
Statistical Analysis 13: Comparison: DIBU Group vs NIBU Group; At one month after primary immunization, the difference between groups (NIBU minus DIBU), in terms of percentage of subjects with pneumococcal antibody concentrations ≥ 0.2 µg/mL were calculated for anti-pneumococccal serotype 5; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 11]; Difference in percentages = -0.64, 98.25% CI 2-sided [-4.63 to 2.92]
Statistical Analysis 14: Comparison: DIBU Group vs NIBU Group; At one month after primary immunization, the difference between groups (NIBU minus DIBU), in terms of percentage of subjects with pneumococcal antibody concentrations ≥ 0.2 µg/mL were calculated for anti-pneumococccal serotype 6B; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 11]; Difference in percentages = -2.38, 98.25% CI 2-sided [-12.02 to 7.22]
Statistical Analysis 15: Comparison: DIBU Group vs NIBU Group; At one month after primary immunization, the difference between groups (NIBU minus DIBU), in terms of percentage of subjects with pneumococcal antibody concentrations ≥ 0.2 µg/mL were calculated for anti-pneumococccal serotype 7F; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 11]; Difference in percentages = 0, 98.25% CI 2-sided [-3.34 to 3.48]
Statistical Analysis 16: Comparison: DIBU Group vs NIBU Group; At one month after primary immunization, the difference between groups (NIBU minus DIBU), in terms of percentage of subjects with pneumococcal antibody concentrations ≥ 0.2 µg/mL were calculated for anti-pneumococccal serotype 9V; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 11]; Difference in percentages = -1.27, 98.25% CI 2-sided [-5.66 to 2.32]
Statistical Analysis 17: Comparison: DIBU Group vs NIBU Group; At one month after primary immunization, the difference between groups (NIBU minus DIBU), in terms of percentage of subjects with pneumococcal antibody concentrations ≥ 0.2 µg/mL were calculated for anti-pneumococccal serotype 14; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 11]; Difference in percentages = 0, 98.25% CI 2-sided [-4.08 to 4.12]
Statistical Analysis 18: Comparison: DIBU Group vs NIBU Group; At one month after primary immunization, the difference between groups (NIBU minus DIBU), in terms of percentage of subjects with pneumococcal antibody concentrations ≥ 0.2 µg/mL were calculated for anti-pneumococccal serotype 18C; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 11]; Difference in percentages = -0.62, 98.25% CI 2-sided [-5.08 to 3.54]
Statistical Analysis 19: Comparison: DIBU Group vs NIBU Group; At one month after primary immunization, the difference between groups (NIBU minus DIBU), in terms of percentage of subjects with pneumococcal antibody concentrations ≥ 0.2 µg/mL were calculated for anti-pneumococccal serotype 19F; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 11]; Difference in percentages = 0.67, 98.25% CI 2-sided [-3.4 to 5.2]
Statistical Analysis 20: Comparison: DIBU Group vs NIBU Group; At one month after primary immunization, the difference between groups (NIBU minus DIBU), in terms of percentage of subjects with pneumococcal antibody concentrations ≥ 0.2 µg/mL were calculated for anti-pneumococccal serotype 23F; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 11]; Difference in percentages = 2.73, 98.25% CI 2-sided [-5.3 to 11.04]

2. Primary Outcome: Antibody Concentrations Against Vaccine Pneumococcal Serotypes
Description: Anti-pneumococcal serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F antibody concentrations have been assessed by 22F-inhibition ELISA, presented as geometric mean concentrations (GMCs) and expressed in micrograms per milliliter (μg/mL). The seropositivity cut-off for the assay was an antibody concentration ≥ 0.05 μg/mL.
Time Frame: One month after primary immunization (At Month 3)
Population: The analysis was performed on the ATP cohort for immunogenicity, which included all evaluable subjects for whom immunogenicity data and assay results for antibodies against at least one study vaccine antigen component after vaccination were available.
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | IIBU Group | DIBU Group | NIBU Group | IPARA Group | DPARA Group | NPARA Group
Number analyzed (Participants) | 154 | 158 | 164 | 55 | 55 | 56
µg/mL
  Anti-1: number analyzed (Participants) | 144 | 155 | 161 | 54 | 51 | 55
  Anti-1 | 1.82 [1.59 to 2.09] | 1.71 [1.49 to 1.95] | 1.9 [1.67 to 2.17] | 1.32 [1.04 to 1.67] | 1.38 [1.09 to 1.74] | 1.95 [1.64 to 2.32]
  Anti-4: number analyzed (Participants) | 146 | 155 | 159 | 55 | 51 | 56
  Anti-4 | 2.25 [1.97 to 2.57] | 2.21 [1.95 to 2.51] | 2.21 [1.96 to 2.5] | 1.57 [1.21 to 2.04] | 1.95 [1.63 to 2.32] | 2.59 [2.07 to 3.24]
  Anti-5: number analyzed (Participants) | 143 | 154 | 157 | 53 | 50 | 54
  Anti-5 | 2.93 [2.58 to 3.33] | 2.39 [2.13 to 2.69] | 2.77 [2.44 to 3.15] | 1.95 [1.53 to 2.48] | 2.36 [1.89 to 2.94] | 3.05 [2.53 to 3.68]
  Anti-6B: number analyzed (Participants) | 144 | 155 | 157 | 53 | 51 | 55
  Anti-6B | 0.67 [0.55 to 0.81] | 0.76 [0.63 to 0.92] | 0.6 [0.49 to 0.72] | 0.49 [0.34 to 0.69] | 0.42 [0.28 to 0.62] | 0.72 [0.51 to 1.02]
  Anti-7F: number analyzed (Participants) | 154 | 157 | 164 | 55 | 55 | 56
  Anti-7F | 2.87 [2.52 to 3.27] | 2.83 [2.52 to 3.17] | 2.77 [2.49 to 3.09] | 2.18 [1.75 to 2.7] | 2.45 [2.01 to 2.99] | 2.95 [2.37 to 3.69]
  Anti-9V: number analyzed (Participants) | 145 | 153 | 157 | 53 | 50 | 54
  Anti-9V | 2.1 [1.81 to 2.42] | 2.01 [1.79 to 2.27] | 2.18 [1.91 to 2.5] | 1.67 [1.3 to 2.13] | 1.82 [1.48 to 2.23] | 2.4 [1.87 to 3.1]
  Anti-14: number analyzed (Participants) | 144 | 154 | 155 | 53 | 50 | 53
  Anti-14 | 4.76 [4.1 to 5.51] | 4.52 [3.91 to 5.21] | 4.77 [4.08 to 5.58] | 3.44 [2.55 to 4.62] | 4.12 [3.21 to 5.29] | 5.17 [4.2 to 6.36]
  Anti-18C: number analyzed (Participants) | 144 | 154 | 157 | 53 | 50 | 54
  Anti-18C | 3.85 [3.23 to 4.6] | 3.8 [3.24 to 4.46] | 4.34 [3.65 to 5.15] | 3.08 [2.29 to 4.15] | 4.08 [3.15 to 5.29] | 4.96 [3.75 to 6.55]
  Anti-19F: number analyzed (Participants) | 145 | 154 | 158 | 53 | 50 | 54
  Anti-19F | 6.11 [5.26 to 7.1] | 5.04 [4.35 to 5.86] | 4.96 [4.22 to 5.83] | 4.95 [3.74 to 6.54] | 5.2 [3.94 to 6.85] | 6.98 [5.48 to 8.88]
  Anti-23F: number analyzed (Participants) | 148 | 158 | 162 | 54 | 53 | 55
  Anti-23F | 1.04 [0.86 to 1.26] | 0.92 [0.76 to 1.11] | 1.07 [0.91 to 1.26] | 0.77 [0.54 to 1.09] | 0.74 [0.51 to 1.08] | 1 [0.73 to 1.36]
Statistical Analysis 1: Comparison: IIBU Group vs NIBU Group; At one month after primary immunization, ELISA Geometric Mean Concentration (GMC) ratios (IIBU over NIBU) were calculated for anti-pneumococcal serotype 1; Test type: Non-Inferiority — A statistically significant decrease in GMC was established if the UL of the two-sided 99.8% CI (adjusted one-sided alpha = 0.11364%) for the GMC ratios (IIBU over NIBU) was below (<) 1 for at least one of the 10 vaccine pneumococcal serotypes; GMC ratio = 0.96, 99.8% CI 2-sided [0.71 to 1.29]
Statistical Analysis 2: Comparison: IIBU Group vs NIBU Group; At one month after primary immunization, ELISA Geometric Mean Concentration (GMC) ratios (IIBU over NIBU) were calculated for anti-pneumococcal serotype 4; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; GMC ratio = 1.02, 99.8% CI 2-sided [0.77 to 1.35]
Statistical Analysis 3: Comparison: IIBU Group vs NIBU Group; At one month after primary immunization, ELISA Geometric Mean Concentration (GMC) ratios (IIBU over NIBU) were calculated for anti-pneumococcal serotype 5; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; GMC ratio = 1.06, 99.8% CI 2-sided [0.8 to 1.41]
Statistical Analysis 4: Comparison: IIBU Group vs NIBU Group; At one month after primary immunization, ELISA Geometric Mean Concentration (GMC) ratios (IIBU over NIBU) were calculated for anti-pneumococcal serotype 6B; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; GMC ratio = 1.12, 99.8% CI 2-sided [0.72 to 1.74]
Statistical Analysis 5: Comparison: IIBU Group vs NIBU Group; At one month after primary immunization, ELISA Geometric Mean Concentration (GMC) ratios (IIBU over NIBU) were calculated for anti-pneumococcal serotype 7F; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; GMC ratio = 1.04, 99.8% CI 2-sided [0.79 to 1.35]
Statistical Analysis 6: Comparison: IIBU Group vs NIBU Group; At one month after primary immunization, ELISA Geometric Mean Concentration (GMC) ratios (IIBU over NIBU) were calculated for anti-pneumococcal serotype 9V; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; GMC ratio = 0.96, 99.8% CI 2-sided [0.7 to 1.31]
Statistical Analysis 7: Comparison: IIBU Group vs NIBU Group; At one month after primary immunization, ELISA Geometric Mean Concentration (GMC) ratios (IIBU over NIBU) were calculated for anti-pneumococcal serotype 14; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; GMC ratio = 1, 99.8% CI 2-sided [0.71 to 1.4]
Statistical Analysis 8: Comparison: IIBU Group vs NIBU Group; At one month after primary immunization, ELISA Geometric Mean Concentration (GMC) ratios (IIBU over NIBU) were calculated for anti-pneumococcal serotype 18C; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; GMC ratio = 0.89, 99.8% CI 2-sided [0.6 to 1.31]
Statistical Analysis 9: Comparison: IIBU Group vs NIBU Group; At one month after primary immunization, ELISA Geometric Mean Concentration (GMC) ratios (IIBU over NIBU) were calculated for anti-pneumococcal serotype 19F; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; GMC ratio = 1.23, 99.8% CI 2-sided [0.87 to 1.75]
Statistical Analysis 10: Comparison: IIBU Group vs NIBU Group; At one month after primary immunization, ELISA Geometric Mean Concentration (GMC) ratios (IIBU over NIBU) were calculated for anti-pneumococcal serotype 23F; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; GMC ratio = 0.97, 99.8% CI 2-sided [0.66 to 1.44]
Statistical Analysis 11: Comparison: DIBU Group vs NIBU Group; At one month after primary immunization, ELISA Geometric Mean Concentration (GMC) ratios (DIBU over NIBU) were calculated for anti-pneumococcal serotype 1; Test type: Non-Inferiority — A statistically significant decrease in GMC was established if the UL of the two-sided 99.8% CI (adjusted one-sided alpha = 0.11364%) for the GMC ratios (DIBU over NIBU) was below (<) 1 for at least one of the 10 vaccine pneumococcal serotypes; GMC ratio = 0.9, 99.8% CI 2-sided [0.67 to 1.21]
Statistical Analysis 12: Comparison: DIBU Group vs NIBU Group; At one month after primary immunization, ELISA Geometric Mean Concentration (GMC) ratios (DIBU over NIBU) were calculated for anti-pneumococcal serotype 4; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 11]; GMC ratio = 1, 99.8% CI 2-sided [0.76 to 1.32]
Statistical Analysis 13: Comparison: DIBU Group vs NIBU Group; At one month after primary immunization, ELISA Geometric Mean Concentration (GMC) ratios (DIBU over NIBU) were calculated for anti-pneumococcal serotype 5; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 11]; GMC ratio = 0.86, 99.8% CI 2-sided [0.66 to 1.14]
Statistical Analysis 14: Comparison: DIBU Group vs NIBU Group; At one month after primary immunization, ELISA Geometric Mean Concentration (GMC) ratios (DIBU over NIBU) were calculated for anti-pneumococcal serotype 6B; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 11]; GMC ratio = 1.28, 99.8% CI 2-sided [0.83 to 1.97]
Statistical Analysis 15: Comparison: DIBU Group vs NIBU Group; At one month after primary immunization, ELISA Geometric Mean Concentration (GMC) ratios (DIBU over NIBU) were calculated for anti-pneumococcal serotype 7F; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 11]; GMC ratio = 1.02, 99.8% CI 2-sided [0.8 to 1.31]
Statistical Analysis 16: Comparison: DIBU Group vs NIBU Group; At one month after primary immunization, ELISA Geometric Mean Concentration (GMC) ratios (DIBU over NIBU) were calculated for anti-pneumococcal serotype 9V; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 11]; GMC ratio = 0.92, 99.8% CI 2-sided [0.69 to 1.22]
Statistical Analysis 17: Comparison: DIBU Group vs NIBU Group; At one month after primary immunization, ELISA Geometric Mean Concentration (GMC) ratios (DIBU over NIBU) were calculated for anti-pneumococcal serotype 14; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 11]; GMC ratio = 0.95, 99.8% CI 2-sided [0.68 to 1.32]
Statistical Analysis 18: Comparison: DIBU Group vs NIBU Group; At one month after primary immunization, ELISA Geometric Mean Concentration (GMC) ratios (DIBU over NIBU) were calculated for anti-pneumococcal serotype 18C; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 11]; GMC ratio = 0.88, 99.8% CI 2-sided [0.6 to 1.27]
Statistical Analysis 19: Comparison: DIBU Group vs NIBU Group; At one month after primary immunization, ELISA Geometric Mean Concentration (GMC) ratios (DIBU over NIBU) were calculated for anti-pneumococcal serotype 19F; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 11]; GMC ratio = 1.02, 99.8% CI 2-sided [0.72 to 1.44]
Statistical Analysis 20: Comparison: DIBU Group vs NIBU Group; At one month after primary immunization, ELISA Geometric Mean Concentration (GMC) ratios (DIBU over NIBU) were calculated for anti-pneumococcal serotype 23F; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 11]; GMC ratio = 0.86, 99.8% CI 2-sided [0.58 to 1.27]

3. Primary Outcome: Antibody Concentrations Against Protein D (Anti-PD)
Description: Anti-PD antibody concentrations were presented as geometric mean concentrations (GMCs), expressed in ELISA units (EL.U) per milliliter (EL.U/mL). The seropositivity cut-off of the assay was an antibody concentration ≥ 100 EL.U/mL.
Time Frame: One month after primary immunization (At Month 3)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | IIBU Group | DIBU Group | NIBU Group | IPARA Group | DPARA Group | NPARA Group
Number analyzed (Participants) | 150 | 158 | 164 | 54 | 53 | 54
EL.U/mL | 1461.3 [1267.4 to 1684.8] | 1353.1 [1191.3 to 1537] | 1557.7 [1355.4 to 1790.3] | 1109.6 [876.9 to 1404.1] | 1348.6 [1048.2 to 1734.9] | 1667.9 [1401.9 to 1984.4]
Statistical Analysis 1: Comparison: IIBU Group vs NIBU Group; At one month after primary immunization, ELISA Geometric Mean Concentration (GMC) ratios (IIBU over NIBU) were calculated for anti-Protein D (anti-PD) antibody; Test type: Non-Inferiority — A statistically significant decrease in GMC was established if the UL of the two-sided 99.8% CI (adjusted one-sided alpha = 0.11364%) for the GMC ratios (IIBU over NIBU) was below (<) 1 for protein D; GMC ratio = 0.94, 99.8% CI 2-sided [0.69 to 1.28]
Statistical Analysis 2: Comparison: DIBU Group vs NIBU Group; At one month after primary immunization, ELISA Geometric Mean Concentration (GMC) ratios (DIBU over NIBU) were calculated for anti-Protein D (anti-PD) antibody; Test type: Non-Inferiority — A statistically significant decrease in GMC was established if the UL of the two-sided 99.8% CI (adjusted one-sided alpha = 0.11364%) for the GMC ratios (DIBU over NIBU) was below (<) 1 for protein D; GMC ratio = 0.87, 99.8% CI 2-sided [0.64 to 1.17]

4. Secondary Outcome: Antibody Concentrations Against Cross-reactive Pneumococcal Serotypes 6A and 19A
Description: Anti-pneumococcal serotype 6A and 19A antibody concentrations have been assessed by 22F-inhibition ELISA, presented as geometric mean concentrations (GMCs) and expressed in micrograms per milliliter (μg/mL). The seropositivity cut-off for the assay was an antibody concentration ≥ 0.05 μg/mL.
Time Frame: One month after primary immunization (At Month 3)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | IIBU Group | DIBU Group | NIBU Group | IPARA Group | DPARA Group | NPARA Group
Number analyzed (Participants) | 147 | 152 | 157 | 53 | 50 | 53
μg/mL
  Anti-6A | 0.17 [0.14 to 0.21] | 0.18 [0.15 to 0.23] | 0.15 [0.12 to 0.19] | 0.11 [0.08 to 0.16] | 0.12 [0.08 to 0.17] | 0.19 [0.13 to 0.27]
  Anti-19A: number analyzed (Participants) | 145 | 152 | 157 | 53 | 50 | 53
  Anti-19A | 0.23 [0.18 to 0.28] | 0.2 [0.16 to 0.25] | 0.16 [0.13 to 0.19] | 0.15 [0.11 to 0.22] | 0.17 [0.12 to 0.25] | 0.25 [0.17 to 0.36]

5. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms
Description: Solicited local symptoms assessed were pain, redness and swelling. Any = incidence of any local symptom regardless of intensity grade. Grade 3 pain = cried when limb was moved/spontaneously painful. Grade 3 redness/swelling = redness/swelling above 30 millimeters (mm).
Time Frame: Within the 4-day (Days 0-3) post-primary vaccination period following each dose and across doses
Population: The analysis was performed on the Total Vaccinated Cohort, which included all vaccinated subjects who received at least one vaccine dose and had the symptoms sheet filled in.
Measure: Count of Participants; unit: Participants
Arm/Group | IIBU Group | DIBU Group | NIBU Group | IPARA Group | DPARA Group | NPARA Group
Number analyzed (Participants) | 197 | 197 | 199 | 70 | 71 | 74
Participants
  Any Pain, Dose 1 | 44 | 48 | 78 | 21 | 28 | 33
  Grade 3 Pain, Dose 1 | 3 | 2 | 8 | 2 | 2 | 7
  Any Redness, Dose 1 | 74 | 52 | 77 | 24 | 19 | 32
  Grade 3 Redness, Dose 1 | 1 | 0 | 1 | 0 | 0 | 0
  Any Swelling, Dose 1 | 29 | 22 | 28 | 10 | 7 | 11
  Grade 3 Swelling, Dose 1 | 1 | 0 | 0 | 0 | 1 | 0
  Any Pain, Dose 2: number analyzed (Participants) | 195 | 197 | 197 | 69 | 71 | 73
  Any Pain, Dose 2 | 60 | 49 | 67 | 19 | 22 | 25
  Grade 3 Pain, Dose 2: number analyzed (Participants) | 195 | 197 | 197 | 69 | 71 | 73
  Grade 3 Pain, Dose 2 | 1 | 2 | 6 | 2 | 0 | 1
  Any Redness, Dose 2: number analyzed (Participants) | 195 | 197 | 197 | 69 | 71 | 73
  Any Redness, Dose 2 | 73 | 59 | 72 | 24 | 23 | 31
  Grade 3 Redness, Dose 2: number analyzed (Participants) | 195 | 197 | 197 | 69 | 71 | 73
  Grade 3 Redness, Dose 2 | 1 | 0 | 0 | 0 | 0 | 2
  Any Swelling, Dose 2: number analyzed (Participants) | 195 | 197 | 197 | 69 | 71 | 73
  Any Swelling, Dose 2 | 31 | 33 | 31 | 10 | 11 | 12
  Grade 3 Swelling, Dose 2: number analyzed (Participants) | 195 | 197 | 197 | 69 | 71 | 73
  Grade 3 Swelling, Dose 2 | 1 | 0 | 0 | 1 | 1 | 2
  Any Pain, Dose 3: number analyzed (Participants) | 194 | 195 | 194 | 69 | 71 | 69
  Any Pain, Dose 3 | 50 | 48 | 52 | 18 | 21 | 22
  Grade 3 Pain, Dose 3: number analyzed (Participants) | 194 | 195 | 194 | 69 | 71 | 69
  Grade 3 Pain, Dose 3 | 2 | 3 | 4 | 1 | 1 | 1
  Any Redness, Dose 3: number analyzed (Participants) | 194 | 195 | 194 | 69 | 71 | 69
  Any Redness, Dose 3 | 70 | 63 | 56 | 28 | 25 | 27
  Grade 3 Redness, Dose 3: number analyzed (Participants) | 194 | 195 | 194 | 69 | 71 | 69
  Grade 3 Redness, Dose 3 | 2 | 0 | 0 | 0 | 2 | 2
  Any Swelling, Dose 3: number analyzed (Participants) | 194 | 195 | 194 | 69 | 71 | 69
  Any Swelling, Dose 3 | 36 | 32 | 30 | 16 | 12 | 13
  Grade 3 Swelling, Dose 3: number analyzed (Participants) | 194 | 195 | 194 | 69 | 71 | 69
  Grade 3 Swelling, Dose 3 | 1 | 0 | 0 | 0 | 0 | 2
  Any Pain, Across doses | 92 | 76 | 107 | 30 | 37 | 44
  Grade 3 Pain, Across doses | 5 | 7 | 15 | 5 | 3 | 7
  Any Redness, Across doses | 108 | 89 | 105 | 36 | 35 | 46
  Grade 3 Redness, Across doses | 4 | 0 | 1 | 0 | 2 | 2
  Any Swelling, Across doses | 61 | 51 | 57 | 20 | 17 | 19
  Grade 3 Swelling, Across doses | 3 | 0 | 0 | 1 | 1 | 2

6. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms
Description: as for outcome 5
Time Frame: Within the 4-day (Days 0-3) period following booster vaccination
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | IIBU-IIBU Group | IIBU-DIBU Group | IIBU-NIBU Group | DIBU-IIBU Group | DIBU-DIBU Group | DIBU-NIBU Group | NIBU-IIBU Group | NIBU-DIBU Group | NIBU-NIBU Group | IPARA-NPARA Group | DPARA-IPARA Group | NPARA-IPARA Group
Number analyzed (Participants) | 63 | 59 | 59 | 60 | 61 | 59 | 60 | 63 | 61 | 66 | 67 | 64
Participants
  Any Pain | 25 | 22 | 15 | 22 | 16 | 25 | 28 | 32 | 28 | 23 | 24 | 24
  Grade 3 Pain | 0 | 3 | 0 | 2 | 1 | 2 | 4 | 1 | 4 | 4 | 4 | 1
  Any Redness | 27 | 25 | 17 | 23 | 15 | 22 | 23 | 25 | 23 | 23 | 23 | 23
  Grade 3 Redness | 0 | 1 | 0 | 0 | 1 | 0 | 3 | 5 | 0 | 0 | 0 | 2
  Any Swelling | 16 | 16 | 9 | 16 | 6 | 11 | 16 | 18 | 15 | 17 | 12 | 16
  Grade 3 Swelling | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0

7. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms
Description: Solicited general symptoms included drowsiness, irritability, loss of appetite and fever [rectally, greater than or equal to (≥) 38 degrees Celsius (°C)]. Any= incidence of any symptom regardless of intensity grade or relationship to vaccination. Grade 3 drowsiness = drowsiness that interfered with normal activity. Grade 3 irritability = crying that could not be comforted/ prevented normal activity. Grade 3 loss of appetite = not eating at all. Grade 3 fever = fever above (>) 40.0°C. Related = symptom assessed by the investigator as related to the vaccination.
Time Frame: Within the 4-day (Days 0-3) post-primary vaccination period following each dose and across doses
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | IIBU Group | DIBU Group | NIBU Group | IPARA Group | DPARA Group | NPARA Group
Number analyzed (Participants) | 197 | 197 | 199 | 70 | 71 | 74
Participants
  Any Drowsiness, Dose 1 | 71 | 78 | 101 | 33 | 28 | 36
  Grade 3 Drowsiness, Dose 1 | 3 | 3 | 3 | 1 | 0 | 1
  Related Drowsiness, Dose 1 | 42 | 47 | 65 | 20 | 17 | 24
  Any Irritability, Dose 1 | 91 | 83 | 109 | 27 | 34 | 43
  Grade 3 Irritability, Dose 1 | 4 | 3 | 6 | 3 | 1 | 3
  Related Irritability, Dose 1 | 61 | 49 | 76 | 18 | 16 | 27
  Any Loss appetite, Dose 1 | 51 | 54 | 71 | 11 | 19 | 32
  Grade 3 Loss appetite, Dose 1 | 0 | 0 | 0 | 0 | 1 | 1
  Related Loss appetite, Dose 1 | 32 | 35 | 43 | 8 | 11 | 20
  Any Fever, Dose 1 | 81 | 73 | 85 | 8 | 11 | 30
  Grade 3 Fever, Dose 1 | 0 | 0 | 0 | 0 | 0 | 0
  Related Fever, Dose 1 | 58 | 56 | 68 | 6 | 8 | 23
  Any Drowsiness, Dose 2: number analyzed (Participants) | 195 | 197 | 197 | 69 | 71 | 73
  Any Drowsiness, Dose 2 | 64 | 66 | 63 | 28 | 15 | 25
  Grade 3 Drowsiness, Dose 2: number analyzed (Participants) | 195 | 197 | 197 | 69 | 71 | 73
  Grade 3 Drowsiness, Dose 2 | 2 | 0 | 2 | 0 | 0 | 1
  Related Drowsiness, Dose 2: number analyzed (Participants) | 195 | 197 | 197 | 69 | 71 | 73
  Related Drowsiness, Dose 2 | 40 | 41 | 43 | 16 | 12 | 15
  Any Irritability, Dose 2: number analyzed (Participants) | 195 | 197 | 197 | 69 | 71 | 73
  Any Irritability, Dose 2 | 79 | 88 | 89 | 30 | 31 | 37
  Grade 3 Irritability, Dose 2: number analyzed (Participants) | 195 | 197 | 197 | 69 | 71 | 73
  Grade 3 Irritability, Dose 2 | 3 | 5 | 5 | 1 | 1 | 1
  Related Irritability, Dose 2: number analyzed (Participants) | 195 | 197 | 197 | 69 | 71 | 73
  Related Irritability, Dose 2 | 56 | 58 | 64 | 20 | 22 | 25
  Any Loss appetite, Dose 2: number analyzed (Participants) | 195 | 197 | 197 | 69 | 71 | 73
  Any Loss appetite, Dose 2 | 52 | 55 | 47 | 12 | 11 | 22
  Grade 3 Loss appetite, Dose 2: number analyzed (Participants) | 195 | 197 | 197 | 69 | 71 | 73
  Grade 3 Loss appetite, Dose 2 | 0 | 0 | 1 | 0 | 0 | 0
  Related Loss appetite, Dose 2: number analyzed (Participants) | 195 | 197 | 197 | 69 | 71 | 73
  Related Loss appetite, Dose 2 | 37 | 41 | 28 | 7 | 8 | 14
  Any Fever, Dose 2: number analyzed (Participants) | 195 | 197 | 197 | 69 | 71 | 73
  Any Fever, Dose 2 | 76 | 55 | 69 | 14 | 15 | 24
  Grade 3 Fever, Dose 2: number analyzed (Participants) | 195 | 197 | 197 | 69 | 71 | 73
  Grade 3 Fever, Dose 2 | 0 | 0 | 0 | 0 | 0 | 1
  Related Fever, Dose 2: number analyzed (Participants) | 195 | 197 | 197 | 69 | 71 | 73
  Related Fever, Dose 2 | 61 | 49 | 55 | 11 | 10 | 19
  Any Drowsiness, Dose 3: number analyzed (Participants) | 194 | 195 | 194 | 69 | 71 | 69
  Any Drowsiness, Dose 3 | 62 | 50 | 45 | 18 | 8 | 16
  Grade 3 Drowsiness, Dose 3: number analyzed (Participants) | 194 | 195 | 194 | 69 | 71 | 69
  Grade 3 Drowsiness, Dose 3 | 1 | 0 | 0 | 0 | 0 | 0
  Related Drowsiness, Dose 3: number analyzed (Participants) | 194 | 195 | 194 | 69 | 71 | 69
  Related Drowsiness, Dose 3 | 40 | 35 | 30 | 12 | 5 | 11
  Any Irritability, Dose 3: number analyzed (Participants) | 194 | 195 | 194 | 69 | 71 | 69
  Any Irritability, Dose 3 | 74 | 68 | 77 | 17 | 21 | 29
  Grade 3 Irritability, Dose 3: number analyzed (Participants) | 194 | 195 | 194 | 69 | 71 | 69
  Grade 3 Irritability, Dose 3 | 3 | 5 | 2 | 1 | 2 | 0
  Related Irritability, Dose 3: number analyzed (Participants) | 194 | 195 | 194 | 69 | 71 | 69
  Related Irritability, Dose 3 | 48 | 48 | 57 | 10 | 12 | 17
  Any Loss appetite, Dose 3: number analyzed (Participants) | 194 | 195 | 194 | 69 | 71 | 69
  Any Loss appetite, Dose 3 | 42 | 41 | 42 | 9 | 9 | 16
  Grade 3 Loss appetite, Dose 3: number analyzed (Participants) | 194 | 195 | 194 | 69 | 71 | 69
  Grade 3 Loss appetite, Dose 3 | 0 | 1 | 3 | 0 | 0 | 1
  Related Loss appetite, Dose 3: number analyzed (Participants) | 194 | 195 | 194 | 69 | 71 | 69
  Related Loss appetite, Dose 3 | 26 | 30 | 26 | 5 | 7 | 12
  Any Fever, Dose 3: number analyzed (Participants) | 194 | 195 | 194 | 69 | 71 | 69
  Any Fever, Dose 3 | 46 | 31 | 42 | 12 | 7 | 14
  Grade 3 Fever, Dose 3: number analyzed (Participants) | 194 | 195 | 194 | 69 | 71 | 69
  Grade 3 Fever, Dose 3 | 0 | 0 | 0 | 0 | 0 | 0
  Related Fever, Dose 3: number analyzed (Participants) | 194 | 195 | 194 | 69 | 71 | 69
  Related Fever, Dose 3 | 38 | 27 | 35 | 7 | 5 | 12
  Any Drowsiness, Across doses | 115 | 111 | 123 | 40 | 33 | 45
  Grade 3 Drowsiness, Across doses | 6 | 3 | 4 | 1 | 0 | 2
  Related Drowsiness, Across doses | 77 | 72 | 87 | 26 | 22 | 32
  Any Irritability, Across doses | 120 | 121 | 138 | 40 | 43 | 59
  Grade 3 Irritability, Across doses | 10 | 12 | 12 | 4 | 4 | 4
  Related Irritability, Across doses | 86 | 82 | 104 | 28 | 28 | 40
  Any Loss appetite, Across doses | 84 | 98 | 100 | 24 | 24 | 42
  Grade 3 Loss appetite, Across doses | 0 | 1 | 3 | 0 | 1 | 2
  Related Loss appetite, Across doses | 56 | 68 | 64 | 16 | 16 | 30
  Any Fever, Across doses | 121 | 101 | 122 | 23 | 27 | 40
  Grade 3 Fever, Across doses | 0 | 0 | 0 | 0 | 0 | 1
  Related Fever, Across doses | 90 | 84 | 101 | 18 | 18 | 31

8. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms
Description: as for outcome 7
Time Frame: Within the 4-day (Days 0-3) period following booster vaccination
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | IIBU-IIBU Group | IIBU-DIBU Group | IIBU-NIBU Group | DIBU-IIBU Group | DIBU-DIBU Group | DIBU-NIBU Group | NIBU-IIBU Group | NIBU-DIBU Group | NIBU-NIBU Group | IPARA-NPARA Group | DPARA-IPARA Group | NPARA-IPARA Group
Number analyzed (Participants) | 63 | 59 | 59 | 60 | 61 | 59 | 60 | 63 | 61 | 66 | 67 | 64
Participants
  Any Drowsiness | 18 | 18 | 17 | 19 | 9 | 21 | 22 | 24 | 24 | 12 | 16 | 19
  Grade 3 Drowsiness | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0
  Related Drowsiness | 15 | 13 | 13 | 13 | 9 | 17 | 17 | 18 | 21 | 10 | 13 | 16
  Any Irritability | 33 | 27 | 23 | 22 | 26 | 27 | 36 | 33 | 32 | 26 | 22 | 27
  Grade 3 Irritability | 1 | 3 | 1 | 3 | 0 | 3 | 3 | 0 | 3 | 2 | 3 | 0
  Related Irritability | 22 | 18 | 13 | 13 | 20 | 23 | 27 | 26 | 27 | 18 | 20 | 16
  Any Loss of appetite | 14 | 16 | 9 | 12 | 15 | 19 | 21 | 24 | 14 | 9 | 10 | 17
  Grade 3 Loss of appetite | 0 | 0 | 0 | 1 | 1 | 0 | 3 | 0 | 1 | 0 | 1 | 0
  Related Loss of appetite | 11 | 11 | 4 | 9 | 15 | 17 | 19 | 19 | 12 | 8 | 6 | 13
  Any Fever | 22 | 21 | 15 | 19 | 19 | 20 | 20 | 23 | 28 | 21 | 14 | 18
  Grade 3 Fever | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Related Fever | 20 | 17 | 12 | 17 | 18 | 18 | 18 | 19 | 24 | 18 | 13 | 16

9. Secondary Outcome: Number of Subjects With Any Serious Adverse Events (SAEs)
Description: SAEs assessed include medical occurrences that results in death, are life threatening, require hospitalization or prolongation of hospitalization, results in disability/incapacity.
Time Frame: During the entire study period (Month 0 to 10)
Population: The analysis was performed on the Total Vaccinated Cohort (TVC), which included all vaccinated subjects who received at least one vaccine dose.
Measure: Count of Participants; unit: Participants
Arm/Group | IIBU Group | DIBU Group | NIBU Group | IPARA Group | DPARA Group | NPARA Group
Number analyzed (Participants) | 198 | 198 | 199 | 71 | 72 | 74
Participants | 4 | 4 | 2 | 4 | 1 | 0

10. Secondary Outcome: Number of Subjects With Any Unsolicited Adverse Events (AEs)
Description: An unsolicited adverse event is any adverse event (i.e. any untoward medical occurrence in a patient or clinical investigation subject, temporally associated with use of a medicinal product, whether or not considered related to the medicinal product) reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms.
Time Frame: Within 31-days (Day 0-30) following each primary vaccination dose
Population: The analysis was performed on the Total Vaccinated Cohort, which included all vaccinated subjects who received at least one vaccine dose.
Measure: Count of Participants; unit: Participants
Arm/Group | IIBU Group | DIBU Group | NIBU Group | IPARA Group | DPARA Group | NPARA Group
Number analyzed (Participants) | 198 | 198 | 199 | 71 | 72 | 74
Participants | 28 | 33 | 35 | 16 | 4 | 13

11. Secondary Outcome: Number of Subjects With Any Unsolicited Adverse Events (AEs)
Description: as for outcome 10
Time Frame: Within 31-days (Day 0-30) following booster vaccination
Population: as for outcome 10
Measure: Number; unit: Subjects
Arm/Group | IIBU-IIBU Group | IIBU-DIBU Group | IIBU-NIBU Group | DIBU-IIBU Group | DIBU-DIBU Group | DIBU-NIBU Group | NIBU-IIBU Group | NIBU-DIBU Group | NIBU-NIBU Group | IPARA-NPARA Group | DPARA-IPARA Group | NPARA-IPARA Group
Number analyzed (Participants) | 64 | 60 | 63 | 63 | 63 | 63 | 63 | 65 | 62 | 67 | 68 | 67
Subjects | 6 | 6 | 2 | 3 | 3 | 4 | 6 | 6 | 3 | 4 | 0 | 2

12. Secondary Outcome: Antibody Concentrations Against Vaccine Pneumococcal Serotypes
Description: Anti- pneumococcal serotypes 1, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F and 23F antibody concentrations have been assessed by 22F-inhibition ELISA, presented as geometric mean concentrations (GMCs) and expressed in micrograms per milliliter (μg/mL). The seropositivity cut-off for the assay was an antibody concentration greater than or equal to (≥) 0.05 μg/mL.
Time Frame: Prior to (Month 9) and one month after booster vaccination (Month 10)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | IIBU-IIBU Group | IIBU-DIBU Group | IIBU-NIBU Group | DIBU-IIBU Group | DIBU-DIBU Group | DIBU-NIBU Group | NIBU-IIBU Group | NIBU-DIBU Group | NIBU-NIBU Group | IPARA-NPARA Group | DPARA-IPARA Group | NPARA-IPARA Group
Number analyzed (Participants) | 50 | 46 | 42 | 48 | 48 | 47 | 46 | 47 | 46 | 50 | 47 | 48
μg/mL
  Anti-1, M9: number analyzed (Participants) | 46 | 44 | 40 | 47 | 44 | 44 | 46 | 44 | 45 | 48 | 41 | 44
  Anti-1, M9 | 0.41 [0.31 to 0.54] | 0.36 [0.28 to 0.46] | 0.27 [0.22 to 0.34] | 0.38 [0.28 to 0.53] | 0.42 [0.31 to 0.57] | 0.34 [0.27 to 0.42] | 0.44 [0.34 to 0.58] | 0.38 [0.3 to 0.48] | 0.43 [0.32 to 0.58] | 0.31 [0.24 to 0.4] | 0.3 [0.23 to 0.4] | 0.45 [0.32 to 0.64]
  Anti-1, M10: number analyzed (Participants) | 49 | 46 | 36 | 44 | 48 | 46 | 44 | 45 | 41 | 47 | 44 | 47
  Anti-1, M10 | 2.87 [2.1 to 3.91] | 2.23 [1.57 to 3.17] | 2.39 [1.68 to 3.41] | 2.69 [1.99 to 3.63] | 2.44 [1.78 to 3.33] | 1.87 [1.36 to 2.57] | 2.84 [2.02 to 3.99] | 3.04 [2.38 to 3.88] | 2.84 [2.1 to 3.85] | 1.76 [1.29 to 2.38] | 2.14 [1.59 to 2.89] | 2.84 [2.06 to 3.89]
  Anti-4, M9: number analyzed (Participants) | 47 | 45 | 40 | 47 | 46 | 45 | 46 | 46 | 45 | 47 | 45 | 45
  Anti-4, M9 | 0.71 [0.55 to 0.92] | 0.63 [0.5 to 0.8] | 0.55 [0.44 to 0.69] | 0.63 [0.47 to 0.85] | 0.72 [0.55 to 0.95] | 0.64 [0.49 to 0.83] | 0.72 [0.55 to 0.93] | 0.73 [0.55 to 0.98] | 0.62 [0.47 to 0.82] | 0.52 [0.39 to 0.68] | 0.6 [0.48 to 0.76] | 0.84 [0.64 to 1.11]
  Anti-4, M10: number analyzed (Participants) | 48 | 45 | 36 | 45 | 47 | 46 | 42 | 45 | 41 | 47 | 45 | 47
  Anti-4, M10 | 4.09 [3.2 to 5.22] | 3.65 [2.76 to 4.84] | 3.22 [2.36 to 4.39] | 4.05 [2.99 to 5.5] | 3.63 [2.84 to 4.62] | 3.41 [2.46 to 4.71] | 4.04 [3.05 to 5.36] | 4.08 [3.11 to 5.36] | 4.07 [3.09 to 5.35] | 3.27 [2.51 to 4.25] | 3.31 [2.66 to 4.12] | 4.28 [3.23 to 5.68]
  Anti-5, M9: number analyzed (Participants) | 46 | 44 | 41 | 47 | 45 | 44 | 46 | 45 | 45 | 47 | 45 | 44
  Anti-5, M9 | 0.98 [0.74 to 1.29] | 0.83 [0.66 to 1.05] | 0.76 [0.59 to 0.98] | 0.78 [0.61 to 1] | 0.76 [0.58 to 0.99] | 0.7 [0.57 to 0.86] | 0.83 [0.66 to 1.05] | 0.84 [0.67 to 1.04] | 0.96 [0.76 to 1.23] | 0.59 [0.45 to 0.77] | 0.72 [0.57 to 0.91] | 0.85 [0.62 to 1.17]
  Anti-5, M10: number analyzed (Participants) | 48 | 45 | 36 | 44 | 48 | 46 | 43 | 45 | 41 | 47 | 45 | 47
  Anti-5, M10 | 4.5 [3.45 to 5.88] | 3.9 [2.95 to 5.16] | 4.11 [2.91 to 5.81] | 3.42 [2.62 to 4.46] | 3.33 [2.56 to 4.33] | 3.37 [2.46 to 4.6] | 4.21 [3.03 to 5.86] | 3.92 [3.06 to 5.01] | 4.48 [3.48 to 5.77] | 2.62 [1.92 to 3.57] | 3.58 [2.74 to 4.69] | 4.33 [3.26 to 5.76]
  Anti-6B, M9: number analyzed (Participants) | 49 | 45 | 41 | 48 | 48 | 47 | 46 | 46 | 45 | 50 | 47 | 45
  Anti-6B, M9 | 0.63 [0.48 to 0.82] | 0.44 [0.31 to 0.61] | 0.54 [0.4 to 0.72] | 0.55 [0.4 to 0.77] | 0.62 [0.48 to 0.8] | 0.6 [0.45 to 0.8] | 0.56 [0.42 to 0.75] | 0.58 [0.43 to 0.78] | 0.67 [0.51 to 0.87] | 0.43 [0.33 to 0.56] | 0.43 [0.33 to 0.57] | 0.61 [0.49 to 0.76]
  Anti-6B M10: number analyzed (Participants) | 49 | 45 | 36 | 45 | 48 | 47 | 44 | 46 | 42 | 48 | 46 | 47
  Anti-6B M10 | 2.75 [2.16 to 3.48] | 1.97 [1.41 to 2.74] | 2.43 [1.85 to 3.19] | 2.13 [1.64 to 2.76] | 2.18 [1.69 to 2.81] | 1.52 [0.98 to 2.34] | 2.16 [1.47 to 3.18] | 2.32 [1.6 to 3.36] | 2.51 [1.96 to 3.22] | 1.74 [1.23 to 2.45] | 1.84 [1.36 to 2.49] | 2.29 [1.79 to 2.91]
  Anti-7F, M9: number analyzed (Participants) | 47 | 43 | 41 | 47 | 46 | 45 | 46 | 45 | 44 | 49 | 43 | 46
  Anti-7F, M9 | 1.33 [1.07 to 1.64] | 0.96 [0.75 to 1.23] | 0.89 [0.74 to 1.07] | 1.08 [0.8 to 1.46] | 1.1 [0.9 to 1.35] | 1.09 [0.89 to 1.34] | 1.07 [0.89 to 1.29] | 1.31 [1.02 to 1.67] | 1.11 [0.83 to 1.49] | 0.84 [0.67 to 1.06] | 0.98 [0.79 to 1.22] | 0.97 [0.76 to 1.24]
  Anti-7F M10: number analyzed (Participants) | 48 | 45 | 36 | 44 | 48 | 47 | 42 | 45 | 41 | 47 | 45 | 47
  Anti-7F M10 | 5.75 [4.59 to 7.21] | 4.2 [3.33 to 5.31] | 4.2 [3.24 to 5.46] | 4.96 [3.77 to 6.54] | 4.36 [3.35 to 5.66] | 3.93 [3.04 to 5.08] | 5.43 [4.13 to 7.14] | 5.55 [4.38 to 7.04] | 4.93 [3.64 to 6.69] | 3.89 [2.98 to 5.1] | 4.63 [3.56 to 6.04] | 4.52 [3.31 to 6.16]
  Anti-9V, M9: number analyzed (Participants) | 48 | 45 | 42 | 47 | 47 | 46 | 46 | 46 | 45 | 50 | 47 | 48
  Anti-9V, M9 | 1.07 [0.82 to 1.39] | 0.83 [0.67 to 1.02] | 0.83 [0.67 to 1.03] | 1.03 [0.79 to 1.36] | 1.03 [0.81 to 1.3] | 0.93 [0.76 to 1.14] | 1.09 [0.83 to 1.44] | 0.92 [0.76 to 1.12] | 1.09 [0.82 to 1.46] | 0.74 [0.58 to 0.95] | 0.93 [0.76 to 1.14] | 0.97 [0.73 to 1.28]
  Anti-9V M10: number analyzed (Participants) | 49 | 46 | 36 | 45 | 48 | 47 | 43 | 47 | 42 | 48 | 46 | 48
  Anti-9V M10 | 4.46 [3.35 to 5.93] | 3.3 [2.47 to 4.41] | 3.94 [2.8 to 5.54] | 3.47 [2.76 to 4.36] | 3.16 [2.39 to 4.17] | 3.07 [2.32 to 4.07] | 4.07 [3 to 5.52] | 3.88 [3.09 to 4.87] | 4.05 [3.18 to 5.15] | 3.11 [2.36 to 4.09] | 3.49 [2.68 to 4.56] | 3.9 [2.86 to 5.3]
  Anti-14, M9: number analyzed (Participants) | 47 | 44 | 41 | 47 | 46 | 46 | 46 | 46 | 45 | 49 | 44 | 46
  Anti-14, M9 | 1.76 [1.23 to 2.51] | 1.74 [1.25 to 2.41] | 1.06 [0.71 to 1.57] | 1.31 [0.99 to 1.74] | 1.7 [1.18 to 2.44] | 1.73 [1.29 to 2.33] | 1.6 [1.06 to 2.39] | 1.93 [1.47 to 2.53] | 1.95 [1.28 to 2.95] | 1.18 [0.85 to 1.64] | 1.53 [1.08 to 2.16] | 1.86 [1.38 to 2.52]
  Anti-14 M10: number analyzed (Participants) | 49 | 46 | 38 | 45 | 48 | 47 | 44 | 46 | 43 | 50 | 47 | 47
  Anti-14 M10 | 6.02 [4.47 to 8.12] | 5.62 [3.99 to 7.92] | 5.16 [3.61 to 7.36] | 4.54 [3.45 to 5.98] | 5.08 [3.8 to 6.8] | 4.61 [3.37 to 6.3] | 6.03 [4.18 to 8.7] | 6.56 [5.06 to 8.51] | 6.3 [4.45 to 8.92] | 4.72 [3.56 to 6.27] | 5.52 [4.13 to 7.38] | 5.62 [4.23 to 7.48]
  Anti-18C M9: number analyzed (Participants) | 50 | 44 | 41 | 47 | 48 | 46 | 46 | 46 | 46 | 50 | 47 | 47
  Anti-18C M9 | 1.13 [0.88 to 1.47] | 1.03 [0.81 to 1.32] | 0.96 [0.73 to 1.26] | 1.08 [0.82 to 1.41] | 1.1 [0.86 to 1.39] | 1.03 [0.8 to 1.31] | 1.12 [0.87 to 1.43] | 1.39 [1.08 to 1.79] | 1.23 [0.93 to 1.63] | 0.91 [0.67 to 1.23] | 1.14 [0.92 to 1.41] | 1.31 [1.01 to 1.69]
  Anti-18C M10: number analyzed (Participants) | 48 | 45 | 38 | 44 | 48 | 47 | 45 | 46 | 42 | 49 | 44 | 47
  Anti-18C M10 | 9.35 [7.13 to 12.25] | 8.06 [5.93 to 10.96] | 7.78 [5.53 to 10.93] | 8.23 [6.37 to 10.65] | 7.16 [5.41 to 9.46] | 7.1 [5.33 to 9.46] | 7.15 [5.13 to 9.96] | 11.29 [7.96 to 16] | 8.68 [6.41 to 11.75] | 6.18 [4.65 to 8.2] | 8.66 [6.76 to 11.09] | 8.17 [5.8 to 11.52]
  Anti-19F M9: number analyzed (Participants) | 46 | 44 | 40 | 46 | 46 | 44 | 46 | 45 | 45 | 48 | 45 | 45
  Anti-19F M9 | 1.94 [1.46 to 2.57] | 1.66 [1.28 to 2.17] | 1.72 [1.23 to 2.39] | 1.58 [1.14 to 2.19] | 1.54 [1.09 to 2.19] | 1.38 [1.09 to 1.75] | 1.25 [0.96 to 1.63] | 1.7 [1.27 to 2.26] | 1.9 [1.38 to 2.62] | 1.56 [1.14 to 2.13] | 1.51 [1.15 to 2] | 1.72 [1.31 to 2.27]
  Anti-19F M10: number analyzed (Participants) | 49 | 45 | 36 | 45 | 48 | 46 | 44 | 45 | 41 | 47 | 44 | 47
  Anti-19F M10 | 6.9 [4.89 to 9.72] | 6.64 [5.17 to 8.54] | 6.91 [4.88 to 9.77] | 5.35 [3.84 to 7.47] | 5.27 [3.64 to 7.64] | 5.57 [4.14 to 7.51] | 5.24 [3.66 to 7.49] | 7.26 [5.28 to 9.97] | 7.34 [5.55 to 9.73] | 5.94 [4.43 to 7.97] | 5.54 [3.88 to 7.93] | 6.66 [4.92 to 9.01]
  Anti-23F M9: number analyzed (Participants) | 48 | 43 | 41 | 47 | 46 | 45 | 46 | 46 | 45 | 49 | 45 | 46
  Anti-23F M9 | 0.65 [0.45 to 0.94] | 0.64 [0.52 to 0.79] | 0.41 [0.28 to 0.58] | 0.55 [0.39 to 0.77] | 0.5 [0.34 to 0.72] | 0.65 [0.5 to 0.84] | 0.61 [0.45 to 0.81] | 0.69 [0.51 to 0.92] | 0.58 [0.43 to 0.79] | 0.47 [0.34 to 0.65] | 0.43 [0.3 to 0.62] | 0.52 [0.37 to 0.74]
  Anti-23F M10: number analyzed (Participants) | 48 | 45 | 35 | 44 | 47 | 46 | 43 | 45 | 41 | 47 | 44 | 47
  Anti-23F M10 | 3.72 [2.6 to 5.33] | 3.08 [2.25 to 4.21] | 2.59 [1.63 to 4.11] | 2.93 [2.05 to 4.19] | 2.16 [1.4 to 3.33] | 2.74 [2.06 to 3.65] | 3.12 [2.17 to 4.48] | 3.17 [2.34 to 4.31] | 3.33 [2.36 to 4.7] | 2.5 [1.76 to 3.56] | 2.53 [1.74 to 3.68] | 3.15 [2.31 to 4.3]
  Anti-6A, M9: number analyzed (Participants) | 46 | 43 | 42 | 47 | 47 | 45 | 46 | 45 | 45 | 48 | 45 | 44
  Anti-6A, M9 | 0.31 [0.21 to 0.46] | 0.18 [0.12 to 0.27] | 0.25 [0.17 to 0.37] | 0.26 [0.18 to 0.39] | 0.32 [0.23 to 0.43] | 0.32 [0.21 to 0.49] | 0.26 [0.17 to 0.4] | 0.28 [0.19 to 0.43] | 0.34 [0.24 to 0.49] | 0.19 [0.13 to 0.27] | 0.22 [0.16 to 0.31] | 0.24 [0.17 to 0.35]
  Anti-6A M10: number analyzed (Participants) | 49 | 46 | 36 | 45 | 48 | 47 | 44 | 46 | 41 | 49 | 47 | 47
  Anti-6A M10 | 1.36 [0.93 to 1.97] | 0.86 [0.56 to 1.34] | 1.14 [0.72 to 1.79] | 0.89 [0.57 to 1.39] | 1.09 [0.78 to 1.54] | 0.74 [0.49 to 1.12] | 1.03 [0.61 to 1.74] | 0.99 [0.66 to 1.48] | 1.4 [0.97 to 2.01] | 0.81 [0.53 to 1.23] | 0.87 [0.59 to 1.29] | 0.98 [0.67 to 1.43]
  Anti-19A M9: number analyzed (Participants) | 47 | 44 | 41 | 46 | 45 | 45 | 46 | 45 | 45 | 48 | 44 | 45
  Anti-19A M9 | 0.28 [0.19 to 0.42] | 0.23 [0.16 to 0.32] | 0.22 [0.15 to 0.32] | 0.24 [0.16 to 0.36] | 0.2 [0.14 to 0.3] | 0.24 [0.17 to 0.33] | 0.15 [0.11 to 0.2] | 0.2 [0.14 to 0.3] | 0.28 [0.19 to 0.4] | 0.21 [0.15 to 0.3] | 0.19 [0.13 to 0.28] | 0.24 [0.16 to 0.36]
  Anti-19A M10: number analyzed (Participants) | 49 | 45 | 35 | 44 | 47 | 46 | 43 | 45 | 41 | 47 | 44 | 47
  Anti-19A M10 | 1.11 [0.67 to 1.83] | 1.1 [0.78 to 1.56] | 1.05 [0.66 to 1.69] | 0.75 [0.48 to 1.15] | 0.66 [0.4 to 1.1] | 0.95 [0.61 to 1.48] | 0.67 [0.43 to 1.04] | 0.93 [0.58 to 1.47] | 0.97 [0.61 to 1.53] | 0.74 [0.49 to 1.1] | 0.63 [0.37 to 1.09] | 1.11 [0.71 to 1.74]

13. Secondary Outcome: Opsonophagocytic Activity (OPA) Titers Against Vaccine Pneumococcal Serotypes
Description: OPA titers against pneumococcal serotypes 1, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F and 23F (Opsono-1, -4, -5, -6A, -6B, -7F, -9V, -14, -18C, -19A, -19F and -23F) were presented as geometric mean titers (GMTs). The seropositivity cut-off for the assay was an antibody titer ≥ 8.
Time Frame: One month after primary immunization (Month 3)
Population: The analysis was performed on the ATP cohort for immunogenicity, which included all evaluable subjects for whom immunogenicity data and assay results or antibodies against at least one study vaccine antigen component after vaccination were available.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | IIBU Group | DIBU Group | NIBU Group | IPARA Group | DPARA Group | NPARA Group
Number analyzed (Participants) | 20 | 16 | 21 | 9 | 13 | 8
Titers
  OPSONO-1: number analyzed (Participants) | 20 | 16 | 21 | 9 | 12 | 8
  OPSONO-1 | 69.4 [26.5 to 182] | 67.9 [28.9 to 159.6] | 75.9 [32.5 to 177] | 23 [6.1 to 86.8] | 94 [31.8 to 277.8] | 64.4 [12.9 to 320.8]
  OPSONO-4 | 1311 [848.8 to 2024.8] | 1172.3 [639.7 to 2148.3] | 1027.7 [573 to 1843.1] | 684.8 [211.7 to 2215.5] | 1712.4 [857 to 3421.6] | 777.2 [119.2 to 5068.1]
  OPSONO-5 | 86.6 [45 to 167] | 52.4 [28.2 to 97.6] | 74.3 [40.6 to 136.1] | 38.7 [14.5 to 103] | 70.7 [29.8 to 167.7] | 80.8 [16.5 to 395]
  OPSONO-6B: number analyzed (Participants) | 20 | 16 | 19 | 9 | 11 | 7
  OPSONO-6B | 723 [434.8 to 1202.3] | 882.4 [331.1 to 2351.7] | 361.3 [125.7 to 1038.4] | 739.9 [346.5 to 1580] | 140.3 [27.6 to 712.2] | 237.1 [30.5 to 1839.6]
  OPSONO-7F: number analyzed (Participants) | 20 | 16 | 18 | 9 | 13 | 7
  OPSONO-7F | 8827.7 [5905.7 to 13195.4] | 4977.9 [3312.3 to 7481.1] | 6444.8 [3781 to 10985.5] | 8362.7 [4221.1 to 16567.7] | 7306.4 [4248.7 to 12564.7] | 6286.1 [3990.3 to 9902.8]
  OPSONO-9V: number analyzed (Participants) | 20 | 16 | 17 | 9 | 11 | 8
  OPSONO-9V | 3429.2 [2184.2 to 5384] | 4040.4 [1816.6 to 8986.3] | 2744.2 [1307.7 to 5758.7] | 5520.1 [2214.2 to 13762] | 3777.1 [1309.9 to 10891.1] | 2273.2 [1339.4 to 3858.3]
  OPSONO-14: number analyzed (Participants) | 20 | 16 | 21 | 9 | 12 | 8
  OPSONO-14 | 1346.3 [522.8 to 3467] | 1219.7 [551.1 to 2699.6] | 1417.9 [940.6 to 2137.3] | 591.5 [121.6 to 2877.4] | 1780.5 [811.9 to 3905] | 1460.1 [777.2 to 2742.9]
  OPSONO-18C: number analyzed (Participants) | 19 | 15 | 18 | 7 | 11 | 7
  OPSONO-18C | 186.9 [129.5 to 269.8] | 167.6 [67.4 to 417.2] | 135.9 [51.4 to 359.5] | 91.6 [13.7 to 611.6] | 382.7 [136 to 1076.8] | 106 [22.2 to 507.2]
  OPSONO-19F: number analyzed (Participants) | 20 | 16 | 18 | 9 | 11 | 7
  OPSONO-19F | 536.2 [361.9 to 794.5] | 514.8 [346.7 to 764.3] | 267.9 [110.4 to 650.3] | 501.1 [247.4 to 1015.3] | 254.2 [59.1 to 1093.9] | 272.1 [45 to 1646]
  OPSONO-23F: number analyzed (Participants) | 20 | 16 | 20 | 9 | 12 | 8
  OPSONO-23F | 989.8 [298.1 to 3286.3] | 1105.5 [323.9 to 3772.4] | 1296 [473.4 to 3548.1] | 1188.4 [206 to 6855.2] | 723 [137.3 to 3805.9] | 838.4 [111.4 to 6313.2]
  OPSONO-6A: number analyzed (Participants) | 20 | 14 | 18 | 9 | 11 | 7
  OPSONO-6A | 79 [25.5 to 245.4] | 151.1 [27.2 to 838.2] | 26.4 [9 to 77] | 100.7 [21.7 to 466.4] | 34.2 [6.4 to 184.1] | 44.5 [4.8 to 411.3]
  OPSONO-19A: number analyzed (Participants) | 14 | 13 | 11 | 6 | 11 | 4
  OPSONO-19A | 16.6 [4.8 to 57.6] | 46.1 [13.4 to 158.2] | 20.4 [5.3 to 79.2] | 11.2 [2.1 to 59.9] | 39.7 [9.9 to 158.5] | 11.4 [0.4 to 315.8]

14. Secondary Outcome: Opsonophagocytic Activity (OPA) Titers Against Vaccine Pneumococcal Serotypes
Description: OPA titers against pneumococcal serotypes (Opsono-1, -4, -5, -6A, -6B, -7F, -9V, -14, -18C, -19A, -19F and -23F) were presented as geometric mean titers (GMTs). The seropositivity cut-off for the assay was ≥ 8. When the number of subjects in a group for a specific category equals (=) 1, the lower limit and upper limit of the confidence interval that can't be calculated, are filled in with the GMT value (due to system constraint). Placeholder value "99999.9" has been entered when value to be entered in the system was greater than (>) 1.0 E10.
Time Frame: Prior to (Month 9) and one month after booster vaccination (Month 10)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | IIBU-IIBU Group | IIBU-DIBU Group | IIBU-NIBU Group | DIBU-IIBU Group | DIBU-DIBU Group | DIBU-NIBU Group | NIBU-IIBU Group | NIBU-DIBU Group | NIBU-NIBU Group | IPARA-NPARA Group | DPARA-IPARA Group | NPARA-IPARA Group
Number analyzed (Participants) | 6 | 6 | 4 | 5 | 8 | 8 | 9 | 5 | 4 | 9 | 11 | 8
Titers
  OPSONO-1, M9: number analyzed (Participants) | 6 | 6 | 3 | 3 | 8 | 8 | 7 | 4 | 4 | 9 | 10 | 8
  OPSONO-1, M9 | 5.8 [2.2 to 15.3] | 4 [4 to 4] | 4 [4 to 4] | 50.3 [0.1 to 18959.2] | 50.6 [10.3 to 248.5] | 9.9 [2.2 to 44.5] | 7.3 [1.7 to 31.9] | 40.2 [2.5 to 638.5] | 10.7 [0.5 to 242.8] | 6 [2.4 to 15] | 12.2 [4.3 to 34.1] | 15.7 [4.4 to 56.3]
  OPSONO-1, M10: number analyzed (Participants) | 5 | 6 | 4 | 5 | 3 | 5 | 9 | 5 | 4 | 5 | 5 | 7
  OPSONO-1, M10 | 346.2 [96.8 to 1237.9] | 296.3 [31 to 2828.6] | 316.4 [96.8 to 1034.8] | 158 [10.2 to 2438.7] | 248 [67.5 to 911.1] | 344.4 [105.7 to 1122.1] | 388.2 [134.4 to 1121.8] | 546.2 [75.4 to 3956.8] | 627 [37 to 10621.6] | 120.6 [10.8 to 1346.5] | 736.3 [184.7 to 2934.6] | 887.6 [226.3 to 3481.1]
  OPSONO-4, M9: number analyzed (Participants) | 4 | 4 | 2 | 1 | 7 | 7 | 6 | 3 | 4 | 8 | 7 | 6
  OPSONO-4, M9 | 34 [0.7 to 1751.4] | 80.2 [3.1 to 2046.3] | 4 [4 to 4] | 9 [9 to 9] | 407.6 [178.5 to 930.7] | 74.2 [10.1 to 546.3] | 98.1 [13.7 to 703] | 52.4 [4 to 681.7] | 15.2 [2.9 to 80.3] | 25.9 [3 to 227] | 56.3 [7.2 to 442] | 161.8 [14.5 to 1807.7]
  OPSONO-4, M10: number analyzed (Participants) | 5 | 6 | 4 | 5 | 3 | 5 | 9 | 5 | 4 | 5 | 6 | 6
  OPSONO-4, M10 | 928.1 [309.6 to 2781.8] | 865.8 [48.5 to 15451.2] | 2213.4 [438.4 to 11174.3] | 2096.7 [828.7 to 5304.9] | 1037.5 [310.2 to 3469.2] | 1096.7 [266.3 to 4516.1] | 1953.4 [972.9 to 3922.2] | 1149.8 [209.9 to 6297.3] | 1414.1 [738.6 to 2707.3] | 548.3 [15 to 20011.5] | 1885.9 [1047.9 to 3394] | 854.4 [51.9 to 14066.3]
  OPSONO-5, M9: number analyzed (Participants) | 6 | 5 | 3 | 3 | 7 | 6 | 7 | 4 | 4 | 9 | 11 | 8
  OPSONO-5, M9 | 12.9 [4.6 to 36.3] | 9.2 [3.2 to 26.5] | 8.2 [0.4 to 185] | 19 [0.5 to 699.8] | 17.5 [4 to 76] | 10.8 [2.8 to 41.7] | 7.6 [2.6 to 21.8] | 12.7 [1.4 to 114.2] | 9.8 [3.7 to 26] | 5.7 [3.3 to 10.1] | 7.4 [4.5 to 12.3] | 22.2 [6.4 to 77]
  OPSONO-5, M10: number analyzed (Participants) | 4 | 6 | 4 | 5 | 3 | 5 | 9 | 5 | 4 | 5 | 7 | 7
  OPSONO-5, M10 | 131.8 [77.7 to 223.6] | 93.3 [15.5 to 562.2] | 241.7 [19.1 to 3061.6] | 79 [7.6 to 826.1] | 114.1 [17.2 to 758.5] | 165.8 [75.4 to 364.8] | 99.5 [36.2 to 273.8] | 128.9 [16.8 to 989.4] | 184.6 [20.4 to 1671.3] | 42.2 [6.3 to 283] | 125.3 [43.6 to 360.3] | 149.7 [27.8 to 806]
  OPSONO-6B, M9: number analyzed (Participants) | 3 | 4 | 3 | 2 | 5 | 5 | 5 | 2 | 4 | 5 | 9 | 1
  OPSONO-6B, M9 | 96.1 [0.1 to 90019.7] | 237.2 [86.5 to 650.7] | 84.3 [0.1 to 63745.1] | 13.3 [0 to 54806323] | 289.4 [9.8 to 8513.4] | 208.9 [12.9 to 3385.1] | 16.4 [1.2 to 229.5] | 13.7 [0 to 86126942] | 182.5 [18.9 to 1765.4] | 127.7 [6.1 to 2672.4] | 105.6 [22.7 to 492.5] | 239 [239 to 239]
  OPSONO-6B, M10: number analyzed (Participants) | 4 | 3 | 3 | 4 | 3 | 4 | 8 | 4 | 2 | 3 | 6 | 5
  OPSONO-6B, M10 | 745.6 [129.8 to 4282.1] | 606.2 [42 to 8748.2] | 769.1 [98.3 to 6016.6] | 694.2 [296.4 to 1626.1] | 553.1 [61.9 to 4943.5] | 1021.6 [405.4 to 2574.3] | 237.6 [50.1 to 1127.3] | 173.1 [2 to 14809] | 1047.8 [203.5 to 5394.1] | 431.5 [26.4 to 7055.2] | 904.3 [416.8 to 1961.9] | 376.5 [92.7 to 1529.8]
  OPSONO-7F, M9: number analyzed (Participants) | 4 | 6 | 3 | 3 | 6 | 7 | 8 | 5 | 4 | 9 | 11 | 5
  OPSONO-7F, M9 | 2076 [972 to 4433.7] | 1777.3 [826.6 to 3821.5] | 1762.5 [499.8 to 6215] | 1729.9 [44.7 to 66995.8] | 5343.2 [1372.2 to 20805] | 3522.8 [1918.3 to 6469.5] | 2563 [1240.6 to 5295.2] | 1152 [421.9 to 3145.6] | 1263.5 [941.3 to 1696] | 1290.9 [705 to 2363.9] | 2256.2 [1405.5 to 3622] | 1744.7 [1196.4 to 2544.2]
  OPSONO-7F, M10: number analyzed (Participants) | 5 | 5 | 3 | 5 | 3 | 4 | 8 | 4 | 3 | 3 | 5 | 5
  OPSONO-7F, M10 | 16259.9 [3902.8 to 67742.7] | 4591.4 [1411.4 to 14936.5] | 12162.6 [776.4 to 190521.8] | 11741 [6560.1 to 21013.7] | 9941.8 [8127.1 to 12161.8] | 5744.5 [1641 to 20109.7] | 14362.4 [7145.2 to 28869.5] | 3565.8 [921.7 to 13795.9] | 5829.1 [2843 to 11951.8] | 11414.1 [394.1 to 330587.3] | 21670 [6757.9 to 69487.8] | 7567.3 [2674.9 to 21408.2]
  OPSONO-9V, M9: number analyzed (Participants) | 5 | 5 | 3 | 3 | 7 | 8 | 7 | 4 | 4 | 9 | 11 | 7
  OPSONO-9V, M9 | 830 [289.3 to 2381] | 1283.8 [523.1 to 3150.9] | 649.4 [55.7 to 7568.6] | 1302.7 [463.1 to 3664.3] | 1423.6 [322.4 to 6284.8] | 1081.9 [332.8 to 3517.5] | 1075.2 [296.2 to 3903.4] | 282.1 [31.3 to 2546.4] | 1571.3 [115.1 to 21457.3] | 567.4 [200.7 to 1604.5] | 480.9 [277.4 to 833.4] | 738.7 [380.4 to 1434.4]
  OPSONO-9V, M10: number analyzed (Participants) | 5 | 4 | 4 | 5 | 3 | 5 | 8 | 4 | 2 | 4 | 6 | 6
  OPSONO-9V, M10 | 4969 [1397.5 to 17668] | 7041.7 [275.3 to 180111.2] | 4756.1 [1023.5 to 22100.8] | 4190.8 [2825.5 to 6215.9] | 3772.9 [80.6 to 176558.2] | 4970.9 [936.8 to 26377] | 4218.9 [1894.6 to 9394.3] | 2919.8 [474 to 17985] | 8601.7 [382.8 to 193287.2] | 856.6 [128.2 to 5724.3] | 7262.2 [2971.8 to 17746.7] | 1340.1 [362 to 4961.2]
  OPSONO-14, M9: number analyzed (Participants) | 5 | 6 | 2 | 2 | 6 | 6 | 6 | 5 | 4 | 8 | 9 | 5
  OPSONO-14, M9 | 149.2 [9.9 to 2241.1] | 255.1 [16.7 to 3888.7] | 47.2 [0 to 99999.9] | 737.1 [1.4 to 400658.5] | 791.7 [200.6 to 3124.5] | 539.2 [251.1 to 1157.8] | 295 [23.9 to 3647.4] | 255.9 [99.2 to 660.2] | 382.6 [115.3 to 1269.1] | 98.3 [15.8 to 613] | 260.7 [132.9 to 511.3] | 195.4 [12.5 to 3045.4]
  OPSONO-14, M10: number analyzed (Participants) | 5 | 5 | 4 | 5 | 3 | 5 | 8 | 5 | 4 | 5 | 6 | 6
  OPSONO-14, M10 | 1592.9 [687.7 to 3689.5] | 671.4 [14.8 to 30474.3] | 4426.6 [692.4 to 28298.7] | 1507.6 [358 to 6348.6] | 2002 [134.3 to 29839.5] | 1312.4 [226.7 to 7597.8] | 1498.1 [672.9 to 3335.6] | 935.3 [301.9 to 2897.7] | 3817 [1256.3 to 11596.8] | 557.5 [17.8 to 17418.8] | 2288 [761.1 to 6878.7] | 587.5 [42.6 to 8103.2]
  OPSONO-18C, M9: number analyzed (Participants) | 4 | 5 | 2 | 2 | 5 | 5 | 8 | 5 | 4 | 8 | 10 | 6
  OPSONO-18C, M9 | 7.2 [1.1 to 45.6] | 7.2 [1.4 to 35.9] | 4 [4 to 4] | 11.5 [0 to 7631549] | 21.9 [2.3 to 205.5] | 10.9 [3.2 to 37.4] | 31.9 [5.9 to 174] | 9.4 [3.4 to 25.9] | 5.5 [2 to 14.8] | 6.5 [3.1 to 13.6] | 19.1 [6.5 to 56.3] | 14 [2.7 to 71.5]
  OPSONO-18C, M10: number analyzed (Participants) | 5 | 4 | 3 | 5 | 3 | 5 | 8 | 3 | 4 | 4 | 6 | 6
  OPSONO-18C, M10 | 912.9 [365.4 to 2280.6] | 207.3 [2.1 to 20168.5] | 2394.7 [2.7 to 2123879] | 397.3 [71.5 to 2207.5] | 650.6 [82.6 to 5122.3] | 298.1 [14.4 to 6180.8] | 428.6 [155.3 to 1183.2] | 707.9 [6.7 to 74589.3] | 481.3 [128.3 to 1804.6] | 149.9 [2.8 to 8106] | 888.9 [225.5 to 3502.9] | 242.7 [24.7 to 2382.5]
  OPSONO-19F, M9: number analyzed (Participants) | 6 | 6 | 3 | 3 | 5 | 6 | 8 | 5 | 4 | 8 | 10 | 7
  OPSONO-19F, M9 | 63 [10.7 to 370.1] | 32.1 [4.2 to 247.3] | 88.5 [0.7 to 11624.3] | 9.7 [0.2 to 438] | 17.7 [1.4 to 226.2] | 67.8 [19 to 242.3] | 15 [5.7 to 39.2] | 24.2 [5.9 to 98.4] | 53.2 [7.7 to 365.3] | 11 [5 to 24.3] | 42.3 [16.4 to 109.6] | 48.4 [12.9 to 181.2]
  OPSONO-19F, M10: number analyzed (Participants) | 5 | 5 | 3 | 5 | 3 | 5 | 9 | 3 | 3 | 5 | 6 | 7
  OPSONO-19F, M10 | 1112.9 [289.7 to 4274.9] | 330.5 [32.2 to 3390.7] | 2575.2 [120.5 to 55029.6] | 637.1 [262.3 to 1547.9] | 1040.7 [12 to 90618.7] | 1575 [246.7 to 10054.3] | 572.7 [332.3 to 986.9] | 273.9 [0 to 2588316] | 250.6 [70.4 to 892.1] | 163.3 [8.6 to 3091.2] | 1215.3 [222.2 to 6647.8] | 511 [59.2 to 4412.4]
  OPSONO-23F, M9: number analyzed (Participants) | 5 | 5 | 3 | 2 | 6 | 7 | 7 | 3 | 4 | 7 | 9 | 5
  OPSONO-23F, M9 | 27.9 [1 to 771.2] | 132.4 [2.3 to 7484.5] | 22.2 [0 to 35490.8] | 29.7 [0 to 99999.9] | 134 [2.2 to 8194.2] | 396.6 [19.4 to 8113.1] | 499.7 [54.2 to 4605.6] | 30.5 [0 to 190610.3] | 15.6 [1.1 to 212.9] | 89.4 [4.8 to 1668.6] | 274.5 [30.2 to 2491.4] | 37.7 [0.8 to 1716.9]
  OPSONO-23F, M10: number analyzed (Participants) | 5 | 6 | 4 | 5 | 3 | 5 | 9 | 5 | 4 | 4 | 7 | 7
  OPSONO-23F, M10 | 581 [14.5 to 23210.4] | 2381.5 [861.8 to 6581] | 2792.9 [391 to 19949.8] | 2977.7 [687.2 to 12903.5] | 2096.1 [823.2 to 5337.4] | 3530.1 [1606.2 to 7758.5] | 4249.1 [2398 to 7529.2] | 3682.7 [1187 to 11426] | 1464.1 [437.9 to 4895.2] | 297 [2 to 44387.7] | 1436.2 [114.1 to 18085.7] | 875.2 [92.2 to 8311]
  OPSONO-6A, M9: number analyzed (Participants) | 4 | 5 | 3 | 3 | 8 | 7 | 8 | 5 | 4 | 6 | 7 | 7
  OPSONO-6A, M9 | 39.8 [0.6 to 2715.5] | 45.1 [2.8 to 721.4] | 13.4 [0.1 to 2451] | 239.5 [21.3 to 2696.8] | 224.8 [41.3 to 1222.9] | 99 [12.8 to 765.5] | 23.3 [3 to 180.7] | 34.1 [1.5 to 760.2] | 58.3 [1.3 to 2537.6] | 46.7 [5.1 to 428.4] | 84 [11.2 to 631.4] | 24.5 [4.1 to 148.1]
  OPSONO-6A, M10: number analyzed (Participants) | 5 | 6 | 4 | 5 | 3 | 4 | 9 | 5 | 3 | 5 | 5 | 7
  OPSONO-6A, M10 | 183.7 [7.3 to 4625.8] | 125.4 [14 to 1123.6] | 318.4 [160.1 to 632.9] | 581.1 [220.5 to 1531.4] | 74.5 [0.1 to 40934.6] | 169.2 [2.9 to 9717.7] | 98.1 [21 to 458.5] | 106.9 [6.5 to 1749.7] | 120 [0.1 to 185061.8] | 154 [8.4 to 2814.5] | 159.1 [9.9 to 2554.8] | 78.5 [10.4 to 592.3]
  OPSONO-19A, M9: number analyzed (Participants) | 3 | 4 | 2 | 2 | 6 | 3 | 6 | 3 | 4 | 6 | 7 | 2
  OPSONO-19A, M9 | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4] | 7.4 [1.5 to 36.3] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4] | 9.1 [2.5 to 33.5] | 4 [4 to 4]
  OPSONO-19A, M10: number analyzed (Participants) | 2 | 2 | 2 | 3 | 3 | 2 | 7 | 1 | 2 | 3 | 5 | 3
  OPSONO-19A, M10 | 363.7 [0 to 5716540] | 4 [4 to 4] | 21.2 [0 to 99999.9] | 28 [0.4 to 1990.5] | 29.8 [0 to 169123.8] | 325.4 [1.9 to 56037.4] | 125.7 [25.1 to 627.8] | 253 [253 to 253] | 12.8 [0 to 33779569] | 44.3 [0.2 to 11784.5] | 416.5 [108.9 to 1593] | 541.6 [22 to 13332.7]

15. Secondary Outcome: Antibody Concentrations Against Protein D (Anti-PD)
Description: Anti-PD antibody concentrations were presented as geometric mean concentrations (GMCs), expressed in ELISA units per milliliter (EL.U//mL). The seroprotection cut-off for the assay was an antibody concentration ≥ 100 EL.U/mL.
Time Frame: Prior to (Month 9) and one month after booster vaccination (Month 10)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | IIBU-IIBU Group | IIBU-DIBU Group | IIBU-NIBU Group | DIBU-IIBU Group | DIBU-DIBU Group | DIBU-NIBU Group | NIBU-IIBU Group | NIBU-DIBU Group | NIBU-NIBU Group | IPARA-NPARA Group | DPARA-IPARA Group | NPARA-IPARA Group
Number analyzed (Participants) | 49 | 45 | 43 | 48 | 48 | 46 | 47 | 47 | 46 | 50 | 48 | 48
EL.U/mL
  Anti-PD, M9: number analyzed (Participants) | 49 | 44 | 43 | 48 | 47 | 45 | 47 | 45 | 46 | 50 | 46 | 48
  Anti-PD, M9 | 661.6 [517.8 to 845.4] | 660.4 [501.1 to 870.4] | 588.3 [431.8 to 801.5] | 622.9 [472 to 821.9] | 590 [456.3 to 763] | 502 [376.6 to 669.2] | 752.1 [561.2 to 1008] | 555.1 [423.1 to 728.2] | 777.2 [561.4 to 1076] | 446.1 [331.1 to 601] | 525.4 [367.8 to 750.4] | 691.3 [550.1 to 868.8]
  Anti-PD M10: number analyzed (Participants) | 49 | 45 | 41 | 46 | 48 | 46 | 46 | 47 | 43 | 50 | 48 | 48
  Anti-PD M10 | 2069 [1639.7 to 2610.8] | 1980.1 [1484.1 to 2641.8] | 1907.5 [1330.9 to 2733.9] | 1888.7 [1349.3 to 2643.6] | 1664.8 [1283 to 2160.2] | 1540.7 [1108.6 to 2141.2] | 2319.7 [1701.9 to 3161.8] | 1953.1 [1541.5 to 2474.5] | 2285.5 [1724.1 to 3029.7] | 1482.7 [1077.1 to 2040.9] | 1517.3 [1134.5 to 2029.2] | 2082.5 [1634.9 to 2652.5]

16. Secondary Outcome: Antibody Concentrations Against Diphtheria (D) and Tetanus (T) Toxoids
Description: Anti-D and anti-T antibody concentrations were presented as geometric mean concentrations (GMCs) and expressed in international units per milliliter (IU/mL). The seroprotection cut-off for the assay was an antibody concentration ≥ 0.1 IU/mL.
Time Frame: One month after primary immunization (Month 3)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | IIBU Group | DIBU Group | NIBU Group | IPARA Group | DPARA Group | NPARA Group
Number analyzed (Participants) | 137 | 150 | 153 | 50 | 49 | 53
IU/mL
  Anti-D | 3.326 [2.97 to 3.725] | 2.938 [2.651 to 3.257] | 3.132 [2.801 to 3.503] | 3.062 [2.565 to 3.655] | 2.891 [2.324 to 3.597] | 3.457 [2.907 to 4.109]
  Anti-T: number analyzed (Participants) | 137 | 150 | 153 | 49 | 49 | 53
  Anti-T | 3.746 [3.305 to 4.245] | 3.373 [3.043 to 3.738] | 3.961 [3.516 to 4.461] | 2.943 [2.434 to 3.559] | 3.058 [2.545 to 3.676] | 3.762 [3.105 to 4.558]

17. Secondary Outcome: Antibody Concentrations Against Diphteria (D) and Tetanus (T) Toxoids
Description: Anti-D and anti-T antibody concentrations were presented as geometric mean concentrations (GMCs) and expressed in IU/mL. The seroprotection cut-off for the assay was an antibody concentration ≥ 0.1 IU/mL.
Time Frame: Prior to (Month 9) and one month after booster vaccination (Month 10)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | IIBU-IIBU Group | IIBU-DIBU Group | IIBU-NIBU Group | DIBU-IIBU Group | DIBU-DIBU Group | DIBU-NIBU Group | NIBU-IIBU Group | NIBU-DIBU Group | NIBU-NIBU Group | IPARA-NPARA Group | DPARA-IPARA Group | NPARA-IPARA Group
Number analyzed (Participants) | 48 | 44 | 40 | 46 | 46 | 45 | 43 | 45 | 43 | 47 | 44 | 47
IU/mL
  Anti-D, M9: number analyzed (Participants) | 45 | 41 | 40 | 46 | 44 | 43 | 43 | 41 | 43 | 46 | 41 | 44
  Anti-D, M9 | 0.736 [0.556 to 0.975] | 0.593 [0.476 to 0.739] | 0.616 [0.499 to 0.762] | 0.55 [0.439 to 0.69] | 0.581 [0.428 to 0.788] | 0.628 [0.483 to 0.815] | 0.714 [0.581 to 0.876] | 0.627 [0.509 to 0.774] | 0.656 [0.514 to 0.836] | 0.665 [0.552 to 0.8] | 0.546 [0.417 to 0.715] | 0.642 [0.518 to 0.795]
  Anti-D, M10: number analyzed (Participants) | 48 | 44 | 34 | 44 | 46 | 45 | 42 | 45 | 40 | 47 | 44 | 47
  Anti-D, M10 | 7.492 [5.932 to 9.463] | 5.257 [4.033 to 6.853] | 7.57 [5.512 to 10.396] | 5.926 [4.752 to 7.39] | 5.831 [4.642 to 7.324] | 6.486 [4.778 to 8.805] | 7.059 [5.455 to 9.136] | 7.226 [5.872 to 8.892] | 8.206 [6.869 to 9.802] | 7.238 [5.322 to 9.845] | 6.477 [5.069 to 8.277] | 6.749 [4.931 to 9.237]
  Anti-T, M9: number analyzed (Participants) | 44 | 40 | 39 | 46 | 44 | 43 | 43 | 41 | 43 | 46 | 40 | 44
  Anti-T, M9 | 0.838 [0.661 to 1.062] | 0.735 [0.573 to 0.944] | 0.66 [0.519 to 0.839] | 0.681 [0.538 to 0.862] | 0.868 [0.668 to 1.13] | 0.692 [0.531 to 0.901] | 0.843 [0.661 to 1.076] | 0.883 [0.686 to 1.136] | 0.858 [0.671 to 1.097] | 0.666 [0.523 to 0.849] | 0.698 [0.538 to 0.907] | 0.9 [0.707 to 1.146]
  Anti-T, M10: number analyzed (Participants) | 48 | 44 | 34 | 44 | 46 | 45 | 43 | 45 | 40 | 47 | 44 | 46
  Anti-T, M10 | 8.03 [6.347 to 10.159] | 6.887 [5.372 to 8.829] | 7.283 [5.179 to 10.243] | 7.092 [5.734 to 8.772] | 7.269 [5.916 to 8.932] | 6.522 [4.886 to 8.707] | 7.095 [5.32 to 9.461] | 10.8 [8.799 to 13.254] | 9.045 [7.659 to 10.681] | 6.491 [4.93 to 8.546] | 7.431 [5.672 to 9.736] | 7.423 [5.625 to 9.796]

18. Secondary Outcome: Antibody Concentrations Against Pertussis Toxoid (Anti-PT), Filamentous Haemagglutinin (Anti-FHA) and Pertactin (Anti-PRN)
Description: Antibody concentrations assessed were presented as geometric mean concentrations (GMCs) and expressed in ELISA units per milliliter (EL.U/mL). The seropositivity cut-off for the assay was an antibody concentration ≥ 5 EL.U/mL.
Time Frame: One month after primary immunization (Month 3)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | IIBU Group | DIBU Group | NIBU Group | IPARA Group | DPARA Group | NPARA Group
Number analyzed (Participants) | 138 | 149 | 155 | 47 | 48 | 53
EL.U/mL
  Anti-PT: number analyzed (Participants) | 133 | 145 | 147 | 47 | 45 | 53
  Anti-PT | 59.1 [53.7 to 65.1] | 64.2 [58.7 to 70.2] | 65 [59.6 to 71] | 60.4 [51.4 to 71] | 63.1 [52 to 76.6] | 61.5 [53.1 to 71.2]
  Anti-FHA: number analyzed (Participants) | 131 | 143 | 142 | 47 | 45 | 52
  Anti-FHA | 163.1 [147.8 to 180.1] | 171.6 [154.7 to 190.4] | 191.1 [171.1 to 213.5] | 171 [139.8 to 209.2] | 196.5 [163.1 to 236.8] | 168.9 [141.9 to 201]
  Anti-PRN | 103.9 [91.5 to 118] | 114.3 [101 to 129.3] | 118.1 [103.9 to 134.3] | 97.1 [76.7 to 123.1] | 106.2 [83.1 to 135.7] | 114 [95.6 to 136]

19. Secondary Outcome: Antibody Concentrations Against Pertussis Toxoid (Anti-PT), Filamentous Haemagglutinin (Anti-FHA) and Pertactin (Anti-PRN)
Description: as for outcome 18
Time Frame: Prior to (Month 9) and one month after booster vaccination (Month 10)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | IIBU-IIBU Group | IIBU-DIBU Group | IIBU-NIBU Group | DIBU-IIBU Group | DIBU-DIBU Group | DIBU-NIBU Group | NIBU-IIBU Group | NIBU-DIBU Group | NIBU-NIBU Group | IPARA-NPARA Group | DPARA-IPARA Group | NPARA-IPARA Group
Number analyzed (Participants) | 48 | 45 | 40 | 46 | 46 | 45 | 45 | 45 | 44 | 49 | 44 | 47
EL.U/mL
  Anti-PT, M9: number analyzed (Participants) | 44 | 40 | 37 | 44 | 43 | 43 | 43 | 39 | 43 | 45 | 38 | 44
  Anti-PT, M9 | 13.3 [10.8 to 16.3] | 12.8 [11 to 14.9] | 10.5 [8.2 to 13.3] | 14.7 [11.1 to 19.6] | 14.2 [11.4 to 17.8] | 13.6 [11.1 to 16.7] | 12.8 [9.9 to 16.7] | 12 [9.1 to 15.9] | 15.2 [12.4 to 18.5] | 13 [10.6 to 16.1] | 10.8 [8.6 to 13.7] | 14.2 [10.5 to 19.1]
  Anti-PT, M10: number analyzed (Participants) | 48 | 44 | 34 | 44 | 46 | 43 | 41 | 44 | 40 | 46 | 44 | 44
  Anti-PT, M10 | 73.8 [58.9 to 92.5] | 64.4 [50.4 to 82.3] | 56.6 [39.9 to 80.5] | 72.3 [57.7 to 90.6] | 75.5 [59.4 to 95.9] | 74.8 [56.9 to 98.2] | 63.4 [48 to 83.6] | 74.9 [60 to 93.4] | 97.6 [82.5 to 115.5] | 59.4 [46.8 to 75.2] | 66.8 [50.6 to 88.3] | 57 [42.2 to 77.1]
  Anti-FHA, M9: number analyzed (Participants) | 44 | 40 | 37 | 44 | 43 | 39 | 43 | 38 | 42 | 45 | 38 | 43
  Anti-FHA, M9 | 46.1 [36.7 to 57.9] | 42.6 [34.5 to 52.6] | 42.6 [33.3 to 54.5] | 53.8 [40.2 to 72.2] | 59.3 [44.1 to 79.8] | 57.7 [41.7 to 79.9] | 57.9 [42.5 to 78.8] | 45.7 [36.3 to 57.6] | 59.1 [46.4 to 75.1] | 50.8 [42.1 to 61.3] | 48.5 [39.7 to 59.3] | 52.9 [39.1 to 71.7]
  Anti-FHA, M10: number analyzed (Participants) | 48 | 44 | 34 | 44 | 46 | 43 | 41 | 44 | 40 | 46 | 44 | 44
  Anti-FHA, M10 | 308.8 [247.1 to 385.9] | 252.7 [195.1 to 327.4] | 327.2 [240.9 to 444.4] | 359.8 [289.2 to 447.6] | 322.9 [252.2 to 413.4] | 332.7 [250.9 to 441.2] | 312.3 [238.7 to 408.8] | 338.6 [270.3 to 424.3] | 442.8 [370.6 to 529] | 321 [246.5 to 417.9] | 332.9 [258.2 to 429.3] | 294.2 [224.3 to 385.9]
  Anti-PRN, M9: number analyzed (Participants) | 47 | 41 | 40 | 46 | 44 | 44 | 45 | 45 | 44 | 49 | 42 | 45
  Anti-PRN, M9 | 15.7 [11.8 to 21.1] | 16 [12.9 to 19.9] | 18.3 [13.8 to 24.4] | 22.4 [16.5 to 30.5] | 25.1 [18.5 to 34] | 16 [11.6 to 22.1] | 19.4 [13.5 to 27.9] | 18.8 [14.1 to 24.9] | 27.3 [20.9 to 35.7] | 20.1 [14.7 to 27.6] | 19.7 [14.6 to 26.7] | 20.3 [14.3 to 29]
  Anti-PRN, M10: number analyzed (Participants) | 48 | 45 | 34 | 44 | 46 | 45 | 42 | 45 | 40 | 49 | 44 | 47
  Anti-PRN, M10 | 218.6 [162.4 to 294.3] | 173.5 [131 to 229.8] | 225.9 [145.9 to 349.8] | 262.9 [196.5 to 351.7] | 246.2 [182.5 to 332] | 184.3 [122.6 to 277.1] | 226.7 [162.6 to 316.1] | 255.7 [189.9 to 344.3] | 330.4 [263.9 to 413.7] | 205.1 [148.5 to 283.5] | 214.2 [151.8 to 302.3] | 213.6 [151.2 to 301.8]

20. Secondary Outcome: Antibody Concentrations Against Hepatitis B Surface Antigen (HBs)
Description: Antibody concentrations assessed were presented as geometric mean concentrations (GMCs) and expressed in milli-international units per milliliter (mIU/mL). The seroprotection cut-off for the assay was an antibody concentration ≥ 10 mIU/mL.
Time Frame: One month after primary immunization (Month 3)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | IIBU Group | DIBU Group | NIBU Group | IPARA Group | DPARA Group | NPARA Group
Number analyzed (Participants) | 111 | 119 | 120 | 40 | 36 | 44
mIU/mL | 911.85 [719.55 to 1155.56] | 1139.1 [902.93 to 1437.04] | 1245.07 [998.97 to 1551.8] | 934.65 [580.7 to 1504.32] | 674.25 [373.26 to 1217.95] | 1027.79 [719.24 to 1468.7]

21. Secondary Outcome: Antibody Concentrations Against Hepatitis B Surface Antigen
Description: Antibody concentrations assessed were presented as geometric mean concentrations (GMCs) and expressed in mIU/mL. The seroprotection cut-off for the assay was an antibody concentration ≥ 10 mIU/mL.
Time Frame: Prior to (Month 9) and one month after booster vaccination (Month 10)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | IIBU-IIBU Group | IIBU-DIBU Group | IIBU-NIBU Group | DIBU-IIBU Group | DIBU-DIBU Group | DIBU-NIBU Group | NIBU-IIBU Group | NIBU-DIBU Group | NIBU-NIBU Group | IPARA-NPARA Group | DPARA-IPARA Group | NPARA-IPARA Group
Number analyzed (Participants) | 43 | 39 | 30 | 41 | 38 | 40 | 34 | 37 | 40 | 37 | 37 | 36
mIU/mL
  Anti-HBs, M9: number analyzed (Participants) | 34 | 35 | 30 | 34 | 35 | 35 | 34 | 30 | 36 | 33 | 33 | 33
  Anti-HBs, M9 | 197.46 [125.7 to 310.18] | 210.32 [125.47 to 352.56] | 164.33 [98.38 to 274.49] | 136.53 [77.08 to 241.83] | 225.01 [135.08 to 374.83] | 194.51 [128.13 to 295.29] | 226.1 [134.4 to 380.39] | 244.52 [133.36 to 448.35] | 159.79 [96.78 to 263.8] | 128.12 [78.68 to 208.6] | 199.57 [115.04 to 346.22] | 209.27 [121.25 to 361.16]
  Anti-HBs, M10: number analyzed (Participants) | 43 | 39 | 29 | 41 | 38 | 40 | 33 | 37 | 40 | 37 | 37 | 36
  Anti-HBs, M10 | 1949.42 [1220.13 to 3114.61] | 1898.54 [1147.47 to 3141.21] | 1970.6 [1017.24 to 3817.44] | 1685.87 [1012.93 to 2805.87] | 2492.42 [1638.97 to 3790.27] | 2107.75 [1257.97 to 3531.56] | 1851.22 [1033.84 to 3314.85] | 2579.59 [1575.91 to 4222.52] | 3244.33 [2235.34 to 4708.75] | 2078.63 [1261.91 to 3423.92] | 2003.09 [1040.72 to 3855.37] | 2218.23 [1219.17 to 4035.97]

22. Secondary Outcome: Antibody Concentrations Against Polyribosyl-ribitol-phosphate (PRP)
Description: Antibody concentrations assessed were presented as geometric mean concentrations (GMCs) and expressed in micrograms per milliliter (µg/mL). The seroprotection cut-off for the assay was an antibody concentration ≥ 0.15 µg/mL.
Time Frame: One month after primary immunization (Month 3)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | IIBU Group | DIBU Group | NIBU Group | IPARA Group | DPARA Group | NPARA Group
Number analyzed (Participants) | 136 | 147 | 150 | 52 | 47 | 53
µg/mL | 3.994 [3.268 to 4.882] | 3.66 [3.073 to 4.359] | 4.51 [3.753 to 5.419] | 3.29 [2.362 to 4.583] | 4.23 [3.025 to 5.914] | 5.007 [3.69 to 6.793]

23. Secondary Outcome: Antibody Concentrations Against Polyribosyl-ribitol-phosphate (PRP)
Description: Antibody concentrations assessed were presented as geometric mean concentrations (GMCs) and expressed in µg/mL. The seroprotection cut-off for the assay was an antibody concentration ≥ 0.15 µg/mL.
Time Frame: Prior to (Month 9) and one month after booster vaccination (Month 10)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | IIBU-IIBU Group | IIBU-DIBU Group | IIBU-NIBU Group | DIBU-IIBU Group | DIBU-DIBU Group | DIBU-NIBU Group | NIBU-IIBU Group | NIBU-DIBU Group | NIBU-NIBU Group | IPARA-NPARA Group | DPARA-IPARA Group | NPARA-IPARA Group
Number analyzed (Participants) | 48 | 45 | 40 | 46 | 47 | 45 | 45 | 45 | 44 | 47 | 44 | 47
µg/mL
  Anti-PRP, M9: number analyzed (Participants) | 46 | 41 | 40 | 46 | 44 | 44 | 45 | 43 | 44 | 46 | 42 | 44
  Anti-PRP, M9 | 0.878 [0.609 to 1.266] | 0.684 [0.48 to 0.974] | 0.678 [0.436 to 1.055] | 0.824 [0.554 to 1.226] | 0.847 [0.571 to 1.256] | 0.763 [0.51 to 1.141] | 0.798 [0.518 to 1.231] | 0.72 [0.531 to 0.977] | 1.013 [0.689 to 1.491] | 0.696 [0.5 to 0.967] | 0.651 [0.452 to 0.938] | 0.953 [0.655 to 1.386]
  Anti-PRP, M10: number analyzed (Participants) | 48 | 45 | 34 | 44 | 47 | 45 | 41 | 45 | 41 | 47 | 44 | 47
  Anti-PRP, M10 | 21.964 [15.76 to 30.61] | 17.484 [11.592 to 26.37] | 21.277 [12.268 to 36.901] | 20.28 [13.96 to 29.462] | 18.987 [13.365 to 26.973] | 17.544 [11.966 to 25.722] | 20.659 [14.948 to 28.55] | 33.45 [23.717 to 47.176] | 22.083 [14.795 to 32.961] | 16.682 [11.367 to 24.481] | 21.602 [14.406 to 32.392] | 23.277 [16.047 to 33.765]

24. Secondary Outcome: Antibody Titers Against Poliovirus Type 1, 2 and 3
Description: Antibody titers assessed were presented as geometric mean titers (GMTs). The seroprotection cut-off for the assay was a titer ≥ the value of 8.
Time Frame: One month after primary immunization (Month 3)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | IIBU Group | DIBU Group | NIBU Group | IPARA Group | DPARA Group | NPARA Group
Number analyzed (Participants) | 24 | 24 | 24 | 11 | 4 | 9
Titers
  Anti-Polio 1: number analyzed (Participants) | 24 | 24 | 24 | 11 | 4 | 8
  Anti-Polio 1 | 283.4 [175.5 to 457.6] | 252.5 [156.9 to 406.2] | 337 [204.2 to 556.2] | 225.6 [103.2 to 492.8] | 166 [97.9 to 281.4] | 449.3 [127.6 to 1581.7]
  Anti-Polio 2: number analyzed (Participants) | 21 | 24 | 24 | 11 | 4 | 9
  Anti-Polio 2 | 362 [259.1 to 505.9] | 327.4 [196.8 to 544.8] | 378 [234.9 to 608.1] | 240.7 [121.9 to 475.3] | 394.8 [99.5 to 1567.1] | 335.2 [152.8 to 735.2]
  Anti-Polio 3: number analyzed (Participants) | 20 | 23 | 21 | 10 | 4 | 9
  Anti-Polio 3 | 423.2 [255.2 to 701.9] | 351.3 [236.4 to 522.1] | 624.1 [394.5 to 987.4] | 284 [151.3 to 533.3] | 394.8 [153.9 to 1012.5] | 438.6 [142.5 to 1349.8]

25. Secondary Outcome: Antibody Titers Against Poliovirus Type 1, 2 and 3
Description: as for outcome 24
Time Frame: Prior to (Month 9) and one month after booster vaccination (Month 10)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | IIBU-IIBU Group | IIBU-DIBU Group | IIBU-NIBU Group | DIBU-IIBU Group | DIBU-DIBU Group | DIBU-NIBU Group | NIBU-IIBU Group | NIBU-DIBU Group | NIBU-NIBU Group | IPARA-NPARA Group | DPARA-IPARA Group | NPARA-IPARA Group
Number analyzed (Participants) | 8 | 7 | 6 | 8 | 8 | 6 | 8 | 5 | 9 | 10 | 4 | 5
Titers
  Anti-Polio 1, M9: number analyzed (Participants) | 5 | 7 | 6 | 8 | 8 | 4 | 6 | 4 | 7 | 4 | 4 | 4
  Anti-Polio 1, M9 | 56 [15.7 to 200.2] | 85.9 [26.7 to 276.4] | 80.9 [18.7 to 349.8] | 145.7 [59.8 to 354.5] | 45.4 [15.9 to 129.6] | 32.1 [11.8 to 87.3] | 67.1 [12.9 to 348.4] | 53.7 [2.7 to 1083.7] | 141.2 [54.2 to 368] | 53.8 [12.5 to 232] | 128.3 [8.4 to 1971.9] | 117.4 [12.7 to 1084]
  Anti-Polio 1, M10: number analyzed (Participants) | 7 | 4 | 4 | 6 | 5 | 6 | 4 | 1 | 7 | 9 | 3 | 4
  Anti-Polio 1, M10 | 1378.2 [682.4 to 2783.4] | 790.7 [75.3 to 8304.9] | 429.9 [35.6 to 5190.7] | 1824.5 [831.6 to 4003] | 388 [60.4 to 2494.6] | 543.9 [79.4 to 3726.3] | 1217.7 [327.7 to 4525.4] | 4 [4 to 4] | 1075.9 [546.1 to 2119.8] | 1290.1 [455.8 to 3651.2] | 1448.1 [148.5 to 14125.5] | 861.1 [74.6 to 9935]
  Anti-Polio 2, M9: number analyzed (Participants) | 6 | 7 | 5 | 8 | 8 | 2 | 7 | 5 | 7 | 5 | 4 | 5
  Anti-Polio 2, M9 | 120.8 [27 to 540.4] | 60.8 [17.8 to 207] | 48.3 [16.3 to 143.4] | 292.1 [61.3 to 1391.9] | 41.7 [19.6 to 88.5] | 8 [0 to 53461.2] | 134.8 [54.1 to 336.1] | 119.6 [25.8 to 553.9] | 156.1 [65.7 to 371] | 29.7 [10.5 to 83.9] | 139.6 [106 to 183.9] | 168.9 [73.8 to 386.4]
  Anti-Polio 2, M10: number analyzed (Participants) | 7 | 4 | 5 | 7 | 5 | 6 | 4 | 2 | 9 | 10 | 3 | 4
  Anti-Polio 2, M10 | 1949 [844.4 to 4498.6] | 1217.7 [101.3 to 14638.5] | 548.7 [41.2 to 7308] | 2151.9 [715.2 to 6474.4] | 512.5 [131.8 to 1993.2] | 542.4 [41.7 to 7057.5] | 1217.7 [195.5 to 7583] | 434.1 [0 to 999999] | 1393.4 [731.1 to 2655.7] | 2047.9 [1068.3 to 3925.7] | 1625.4 [270.8 to 9756.8] | 1116.6 [126.6 to 9848.8]
  Anti-Polio 3, M9: number analyzed (Participants) | 6 | 7 | 5 | 8 | 8 | 3 | 8 | 4 | 7 | 5 | 4 | 4
  Anti-Polio 3, M9 | 72 [18.9 to 273.5] | 86 [33.8 to 218.9] | 127.8 [30.6 to 534.2] | 205.4 [52.5 to 804.1] | 45.3 [14.2 to 144.4] | 45.2 [19.1 to 106.8] | 70 [31.6 to 155.4] | 139.6 [30.5 to 638.7] | 128 [75.8 to 216.3] | 96.5 [12.3 to 758.1] | 108.1 [62.5 to 186.8] | 69.7 [2.2 to 2175.5]
  Anti-Polio 3, M10: number analyzed (Participants) | 8 | 4 | 4 | 6 | 5 | 6 | 4 | 2 | 8 | 10 | 3 | 1
  Anti-Polio 3, M10 | 861 [363.5 to 2039.4] | 1724.5 [66.3 to 44854.5] | 359.5 [8.4 to 15474.7] | 3649.1 [1721.5 to 7735.1] | 588.1 [44 to 7860.3] | 1152.5 [123.7 to 10737.5] | 558.3 [140.6 to 2216.3] | 724.1 [0 to 999999] | 2233.3 [1122.1 to 4445] | 2195 [889 to 5419.4] | 1625.4 [436.4 to 6054.1] | 2048 [2048 to 2048]

ADVERSE EVENTS:
Time Frame: Solicited local/general symptoms: during the 4-day (Days 0-3) follow-up periods after primary and booster vaccination. Unsolicited AEs: during the 31-day (Days 0-30) follow-up periods after primary and booster vaccination. SAEs: during the entire study period (from Month 0 up to Month 10).
Arm/Group | IIBU Group | DIBU Group | NIBU Group | IPARA Group | DPARA Group | NPARA Group | IIBU-IIBU Group | IIBU-DIBU Group | IIBU-NIBU Group | DIBU-IIBU Group | DIBU-DIBU Group | DIBU-NIBU Group | NIBU-IIBU Group | NIBU-DIBU Group | NIBU-NIBU Group | IPARA-NPARA Group | DPARA-IPARA Group | NPARA-IPARA Group
All-Cause Mortality (participants affected / at risk) | 0/198 | 0/198 | 0/199 | 0/71 | 0/72 | 0/74 | 0/64 | 0/60 | 0/63 | 0/63 | 0/63 | 0/63 | 0/63 | 0/65 | 0/62 | 0/67 | 0/68 | 0/67
Serious Adverse Events (participants affected / at risk) | 4/198 | 4/198 | 2/199 | 4/71 | 1/72 | 0/74 | 0/64 | 1/60 | 0/63 | 0/63 | 0/63 | 0/63 | 0/63 | 1/65 | 0/62 | 1/67 | 0/68 | 0/67
Other Adverse Events (participants affected / at risk) | 181/198 | 171/198 | 186/199 | 60/71 | 61/72 | 73/74 | 44/64 | 41/60 | 34/63 | 43/63 | 41/63 | 42/63 | 50/63 | 51/65 | 45/62 | 43/67 | 45/68 | 45/67
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IIBU Group (N=198) | DIBU Group (N=198) | NIBU Group (N=199) | IPARA Group (N=71) | DPARA Group (N=72) | NPARA Group (N=74) | IIBU-IIBU Group (N=64) | IIBU-DIBU Group (N=60) | IIBU-NIBU Group (N=63) | DIBU-IIBU Group (N=63) | DIBU-DIBU Group (N=63) | DIBU-NIBU Group (N=63) | NIBU-IIBU Group (N=63) | NIBU-DIBU Group (N=65) | NIBU-NIBU Group (N=62) | IPARA-NPARA Group (N=67) | DPARA-IPARA Group (N=68) | NPARA-IPARA Group (N=67)
Accidental poisoning (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Convulsion (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypotonia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rickets (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchiolitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis rotavirus (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Laryngitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Otitis media (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IIBU Group (N=198) | DIBU Group (N=198) | NIBU Group (N=199) | IPARA Group (N=71) | DPARA Group (N=72) | NPARA Group (N=74) | IIBU-IIBU Group (N=64) | IIBU-DIBU Group (N=60) | IIBU-NIBU Group (N=63) | DIBU-IIBU Group (N=63) | DIBU-DIBU Group (N=63) | DIBU-NIBU Group (N=63) | NIBU-IIBU Group (N=63) | NIBU-DIBU Group (N=65) | NIBU-NIBU Group (N=62) | IPARA-NPARA Group (N=67) | DPARA-IPARA Group (N=68) | NPARA-IPARA Group (N=67)
Pain (General disorders) | 92 (154) | 76 (145) | 107 (197) | 30 (58) | 37 (71) | 44 (80) | 25 (25) | 22 (22) | 15 (15) | 22 (22) | 16 (16) | 25 (25) | 28 (28) | 32 (32) | 28 (28) | 23 (23) | 24 (24) | 24 (24)
Pyrexia (General disorders) | 121 (205) | 102 (165) | 123 (200) | 23 (35) | 28 (35) | 40 (68) | 22 (22) | 21 (21) | 15 (15) | 19 (19) | 19 (19) | 20 (20) | 20 (20) | 23 (23) | 28 (28) | 21 (21) | 14 (14) | 18 (18)
Swelling (General disorders) | 61 (96) | 51 (87) | 57 (89) | 20 (36) | 17 (30) | 19 (36) | 16 (16) | 16 (16) | 9 (9) | 16 (16) | 6 (6) | 11 (11) | 16 (16) | 18 (18) | 15 (15) | 17 (17) | 12 (12) | 16 (16)
Nasopharyngitis (Infections and infestations) | 5 (5) | 3 (3) | 3 (4) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 5 (6) | 5 (6) | 10 (14) | 3 (3) | 0 (0) | 3 (4) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 4 (5) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 84 (145) | 98 (150) | 100 (160) | 25 (33) | 24 (39) | 42 (70) | 14 (14) | 16 (16) | 9 (9) | 12 (12) | 15 (15) | 19 (19) | 21 (21) | 24 (24) | 14 (14) | 9 (9) | 10 (10) | 17 (17)
Somnolence (Nervous system disorders) | 115 (197) | 111 (194) | 123 (209) | 40 (79) | 33 (51) | 45 (77) | 18 (18) | 18 (18) | 17 (17) | 19 (19) | 9 (9) | 21 (21) | 22 (22) | 24 (24) | 24 (24) | 12 (12) | 16 (16) | 19 (19)
Irritability (Psychiatric disorders) | 120 (244) | 121 (239) | 138 (275) | 41 (75) | 43 (86) | 59 (109) | 33 (33) | 27 (27) | 23 (23) | 22 (22) | 26 (26) | 27 (27) | 36 (36) | 33 (33) | 32 (32) | 26 (26) | 22 (22) | 27 (27)
Erythema (Skin and subcutaneous tissue disorders) | 108 (217) | 89 (174) | 105 (205) | 36 (76) | 35 (67) | 46 (90) | 27 (27) | 25 (25) | 17 (17) | 23 (23) | 15 (15) | 22 (22) | 23 (23) | 25 (25) | 23 (23) | 23 (23) | 23 (23) | 23 (23)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.